

**Official Title:** A Multicenter, Multinational, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 190 in Patients with CLN2 Disease

NCT Number: NCT02485899

Applicant/MAH: BioMarin Pharmaceutical Inc.

**Version Date:** 17 December 2018



## CLINICAL STUDY PROTOCOL

A Multicenter, Multinational, Extension Study to Evaluate the **Study Title:** 

Long-Term Efficacy and Safety of BMN 190 in Patients with

**CLN2** Disease

**Protocol Number:** 190-202

Cerliponase alfa (BMN 190), recombinant human tripeptidyl **Active Investigational Product:** 

peptidase 1 (rhTPP1)

IND/European Union Drug **Regulating Authorities Clinical** Trials (EudraCT) Number:

IND 122472 / EudraCT 2014-003480-37

CLN2 disease due to tripeptidyl peptidase 1 (TPP1) deficiency **Indication:** 

BioMarin Pharmaceutical Inc.

**Sponsor:** 105 Digital Drive

Novato, CA 94949

Phase 1/2 Extension **Development Phase:** , MD

Sponsor's Responsible Medical

Monitor: Sr. Medical Director, Rare Disease

**Study Design:** Open-label Extension Up to 240 weeks

**Duration of Subject** 

Participation:

Dose:

300 mg BMN 190 every-other-week

Patients with confirmed diagnosis of CLN2, who completed **Study Population:** 

participation in 190-201

3 October 2014 **Date of Original Protocol: Date of Protocol Amendment 1:** 12 August 2015 **Date of Protocol Amendment 2:** 16 November 2015 **Date of Protocol Amendment 3:** 26 February 2016 **Date of Protocol Amendment 4:** 17 March 2017 **Date of Protocol Amendment 5:** 05 May 2017 **Date of Protocol Amendment 6** 17 December 2018

## **Property of BioMarin CONFIDENTIAL**

May not be divulged, published, or otherwise disclosed to others without prior written approval from BioMarin.

This study will be conducted according to the principles of Good Clinical Practice as described in the U.S. Code of Federal Regulations and the International Conference on Harmonisation Guidelines, including the archiving of essential documents.



## CLINICAL STUDY PROTOCOL AMENDMENT SUMMARY

Amendment: 6

Date: 17 December 2018

## SUMMARY OF CHANGES AND RATIONALE

This section provides a numbered list of all significant changes and supporting rationale.

- 1. Updates were made to the immunogenicity assessment section to include serum neutralizing antibodies (NAb) sample collection. This change was made in response to a Regulatory Agency request to evaluate the presence of neutralizing antibodies to BMN 190 in serum. No changes are being made to the frequency or schedule of assessments.
- 2. Added clarification that for subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug.
- 3. Re-classified electroencephalogram (EEG) from the list of safety assessment to efficacy assessments as this test provides information regarding changes in electrical activity in the brain while on study drug, but does not provide safety information used to determine whether dose modification or interruption is warranted.
- 4. Added that central laboratories (or a central reviewer) will be used to evaluate EEG scans in order to standardize review and data presentation, and limit site-associated variability.
- 5. Added CLN2 disease rating scale assessment to the 4-week device safety follow-up visit and 6-month safety follow-up visit in order to ascertain whether there were any functional changes associated with any reported adverse events.
- 6. Added ophthalmology/visual acuity assessment every 12 weeks and optical coherence tomography every 24 weeks in order to provide additional data to supplement the vision domain of the CLN2 rating scale.
- 7. Removed EQ-5D-5L Questionnaire in order to decrease study burden and the determination that the other Quality of Life questionnaires administered may be more relevant to this patient population.



- 8. Frequency of complete physical examination was changed from every 12 weeks to every 48 weeks to decrease burden to the subjects. The frequency of the brief physical exam remains unchanged (every 2 weeks). Assessment of height and body weight has been changed from every 48 weeks to every 24 weeks to permit additional monitoring of growth milestones.
- 9. Added updated information that the material degradation of the ICV device reservoir has occurred after approximately 105 perforations of the ICV device in benchtop testing, and has been observed in clinical trials with approximately 4 years of BMN 190 administration. Access device replacement should be considered prior to 4 years of regular administration of BMN 190; with the decision made on an individual subject level based on the medical judgment of the Investigator.
- 10. Clarified the stopping criteria that subjects with a score of 0 on the combined motor and language components of the Hamburg CLN2 rating scale at two consecutive visits will be discontinued from treatment.
- 11. Clarified that, in the event of a device-related AE where the device and its components should be returned to BioMarin for further testing, the infusion pump does not need to be returned.
- 12. Updated Introduction to reflect interim 96-week results from the ongoing extension study (190-201 and 190-202).
- 13. Administrative changes have been made for consistency and clarity.

Refer to Section 25 for a summary of the amendment revisions.



### 2 SYNOPSIS

| NAME OF COMPANY | SUMMARY TABLE | FOR NATIONAL |
|---|---|---|
| BioMarin Pharmaceutical Inc. | Referring to Part of the | AUTHORITY |
| 105 Digital Drive | Dossier: | <b>USE ONLY:</b> |
| Novato, CA 94949 | | |
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume: Page: Reference: | |
| NAME OF ACTIVE INGREDIENT: | | |
| recombinant human tripeptidyl peptidase 1 | | |

### TITLE OF STUDY:

A Multicenter, Multinational, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 190 in Patients with CLN2 Disease

### PROTOCOL NUMBER:

190-202

#### STUDY SITES:

Approximately 10 centers worldwide

## PHASE OF DEVELOPMENT:

Phase 1/2 Extension

### STUDY RATIONALE:

BMN 190 is a recombinant form of human tripeptidyl peptidase 1 (TPP1), the enzyme deficient in patients with CLN2 disease (also known as classical late-infantile CLN2, cLINCL, or Jansky-Bielschowsky disease), a form of Batten Disease. As an enzyme replacement therapy (ERT), BMN 190, is expected to restore TPP1 enzyme activity. Given the urgent and severe unmet medical need in CLN2 disease and observations in neurologically relevant animal models of CLN2 disease, clinical development of BMN 190 ERT is justified.

Murine and canine models of CLN2 disease (sharing the same genetic and enzymatic defect TPP1 deficiency, as the human disorder) recapitulate the major human clinical signs and pathology, including neuron loss, tremor, ataxia, functional decline, and reduced lifespan. ERT with BMN 190 administered intrathecally or via intracerebroventricular infusion in both models yielded pharmacologically significant benefit. Furthermore, when dosing of BMN 190 started early in life (~2.5 months of age) in the TPP1-null dachshund model, BMN 190 significantly delayed onset of clinical signs, preserved motor and cognitive function, and prolonged life. The better pharmacological response to ERT in this and other animal models, when treatment was started closer to birth, indicates the importance of starting therapy as early in life as possible. There is currently no accepted, standard treatment for CLN2 other than supportive care. Enzyme

There is currently no accepted, standard treatment for CLN2 other than supportive care. Enzyme replacement therapy (ERT) with BMN 190, or recombinant human TPP1 (rhTPP1), is a potential new treatment option for CLN2 patients. BMN 190 is expected to reduce the progressive, pathologic accumulation of lysosomal storage material, and improve the symptoms of disease.

The Phase 1/2 study (190-201) evaluated the efficacy and safety of doses up to 300 mg/every other week (qow) BMN 190 in patients with CLN2. Results from the 190-201 study demonstrated a substantial improvement of the rate of clinical progression in children treated with BMN 190 compared with untreated historical controls. Further, in those children who had received at least

|----------|---------------------|--------|
|----------|---------------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY<br>USE ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume:<br>Page:<br>Reference: | |
| NAME OF ACTIVE INGREDIENT: | | |
| recombinant human tripeptidyl peptidase 1 | . 1 21 | |

48 weeks of BMN 190 dosing, clinical scores stabilized, in contrast to matched historical untreated controls in which decline was rapid and profound in the majority of matches.

The dose and regimen for this study (190-202) are based on the results of the 190-201 study. The rationale for this phase 2 extension study is to provide patients who complete the 190-201 study with the option to continue BMN 190 treatment. The 190-202 study is an open label extension protocol to assess long-term safety and efficacy.

### **OBJECTIVES:**

The primary objective of the study is:

- To evaluate the long-term safety of BMN 190 administration at 300 mg qow in patients with CLN2.
- To assess change in motor and language (ML) subscales of the CLN2 disease rating scale in patients with CLN2 receiving BMN 190 at 300 mg gow.

The secondary objectives of the study are:

- To assess changes in quantitative assessment of MRI.
- To assess change in CLN2 disease scale total score.
- To evaluate quality of life (QoL) with long-term BMN 190 administration.

The exploratory objective of the study is:

- To evaluate age-appropriate developmental milestones with long-term BMN 190 administration.
- To evaluate the impact of treatment on disease-related biomarkers from CSF and blood.

## STUDY DESIGN AND PLAN:

This is a multi-center, multinational, extension study to evaluate BMN 190 treatment in patients with CLN2 who completed 190-201. All patients who have completed 48 weeks in Study 190-201 will be eligible to enroll in Study 190-202.

The Screening period for Study 190-202 will start simultaneously with the Week 47 visit in Study 190-201. Baseline values for Study 190-202 will be recorded at the first infusion, Week 1 Day 1 of Study BMN 190-202, for all patients on active treatment. The first dose of BMN 190 in Study 190-202 (Week 1/Study Day 1) will be given following the Week 49 study assessments in Study 190-201. This study will be open label with all patients continuing on treatment with BMN 190 300 mg gow.

|------------------------------|--------|
|------------------------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY<br>USE ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume: Page: Reference: | |
| NAME OF ACTIVE INGREDIENT: recombinant human tripeptidyl peptidase 1 | | |

Patients will complete safety and efficacy assessments including CSF surveillance labs every 2 weeks, CLN2 disease scales every 8 weeks, clinical laboratory assessments, visual acuity tests, and immunogenicity tests every 12 weeks. MRI, quality of life measures, OCT, EEG, developmental milestones (Denver II), and blood and CSF samples for evaluating disease-related biomarkers will be collected every 24 weeks. Complete physical examination will be performed every 48 weeks. Some patients may experience hypersensitivity reactions, thus prophylactic antihistamine and/or antipyretic may be administered prior to each study drug infusion at the investigator's discretion. To date, there has been no anaphylaxis or anaphylactoid reactions in studies with BMN 190. However, in the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion).

In addition, the investigator must contact the BioMarin medical monitor within 1 business day if any AE is severe (Grade 3 or higher) or serious and requires any of the following:

- infusion interruption, discontinuation, or modification (not due to blocked line)
- administration of IV fluids, steroids, or antihistamines
- administration of oxygen

Before subsequent infusions, the study site investigator and BioMarin medical monitor will discuss the case and agree upon infusion modification or additional premedication, if necessary. Agreed upon dose modifications or introduction of additional premedication should be documented in the Electronic Case Report Forms (eCRFs) and source files.

Patients may withdraw voluntarily from receiving study drug at any time, yet will be encouraged to continue to undergo study assessments. Patients may also withdraw entirely from complete study participation at any time, upon request.

## NUMBER OF PATIENTS PLANNED:

All patients who complete 48 weeks in the 190-201 study may be eligible to enroll.

## DIAGNOSIS AND ALL CRITERIA FOR INCLUSION AND EXCLUSION:

To be eligible for study participation, a patient must meet all of the following inclusion criteria:

• Must have completed 48 weeks in Study 190-201.

|----------|---------------------|--------|
|----------|---------------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY<br>USE ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume:<br>Page:<br>Reference: | |
| <b>NAME OF ACTIVE INGREDIENT:</b> recombinant human tripeptidyl peptidase 1 | | |

- Is willing and able to provide written, signed informed consent. Or, in the case of patients under the age of 18 (or other age as defined by regional law or regulation), provide written assent (if required) and have written informed consent, signed by a legally authorized representative, after the nature of the study has been explained, and prior to performance of research-related procedures.
- Males and females who are of reproductive age should practice true abstinence, defined as no sexual activity, during the study and for 6 months after the study has been completed (or withdrawal from the study). If sexually active and not practicing true abstinence, males and females of reproductive age must use a highly effective method of contraception while participating in the study.
- If female, of childbearing potential, must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests done during the study.

If any of the following exclusion criteria apply, a patient will not be eligible to participate in the study:

- Has had a loss of 3 or more points in the combined motor and language components of the Hamburg CLN2 rating scale between Baseline of Study 190-201 and the Study Completion visit in Study 190-201 and would not benefit from enrolling in the study in the Investigator's discretion.
- Has a score of 0 points on the combined motor and language components of the Hamburg CLN2 rating scale.
- Is pregnant or breastfeeding, at Baseline, or planning to become pregnant (self or partner) at any time during the study.
- Has used any investigational product (other than BMN 190), or investigational medical device, within 30 days prior to Baseline; or is required to use any investigational agent prior to completion of all scheduled study assessments.
- Has a concurrent disease or condition that would interfere with study participation, or pose a safety risk, as determined by the Investigator.
- Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

| BIOMARIN 190-202 Amendment 6 Page | e 8 |
|-----------------------------------|-----|
|-----------------------------------|-----|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY<br>USE ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume:<br>Page:<br>Reference: | |
| NAME OF ACTIVE INGREDIENT: recombinant human tripeptidyl peptidase 1 | | |

### INVESTIGATIONAL PRODUCT, DOSE, ROUTE AND REGIMEN:

All study subjects will be administered BMN 190 300 mg by ICV infusion every other week (preferably in the morning). Fasting for a minimum of 2 hours before each infusion may be considered until the subject's reaction to the study drug is determined. When a feeding tube is used for an overnight feed, the tube may be turned off 2 hours before infusion.

## REFERENCE THERAPY, DOSE, ROUTE AND REGIMEN:

Because practical and ethical concerns preclude contemporaneous or untreated control subjects, comparison will be with historical data from existing CLN2 disease registries.

### **DURATION OF TREATMENT:**

Patients will receive qow ICV infusions of study drug, up to Week 239 or until one of the following occurs: the patient withdraws consent and discontinues from the study; the patient is discontinued from the study at the discretion of the Investigator; the patient enrolls in another study or registry; or the study is terminated.

### **CRITERIA FOR EVALUATION:**

### Safety:

- AEs and concomitant medication
- routine clinical laboratory tests (hematology, chemistry, and urinalysis)
- routine CSF surveillance (cell, count, protein, and glucose)
- vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], heart rate, respiration rate, and temperature)
- physical examination (including height)
- electrocardiogram (ECG), 3- or 5-lead, 12-lead
- immunogenicity, includes anti-BMN 190 total antibodies (TAb) and neutralizing antibodies (Nab) in CSF; TAb, NAb, total IgE, and drug-specific IgE in serum

# Efficacy:

- CLN2 disease rating scales with videotaping
- Total cortical grey matter volume
- Quality of Life surveys
- Developmental assessments
- Disease-related biomarkers
- EEG, standard awake
- Assessments of visual acuity
- Optical coherence tomography

|------------------------------|--------|
|------------------------------|--------|

| NAME OF COMPANY BioMarin Pharmaceutical Inc. 105 Digital Drive Novato, CA 94949 | SUMMARY TABLE Referring to Part of the Dossier: | FOR NATIONAL<br>AUTHORITY<br>USE ONLY: |
|---|---|---|
| NAME OF FINISHED PRODUCT:<br>Cerliponase alfa (BMN 190) | Volume: Page: Reference: | |
| NAME OF ACTIVE INGREDIENT: recombinant human tripeptidyl peptidase 1 | | |

# Immunogenicity:

• TAb and NAb in CSF; TAb, NAb, total IgE, and drug-specific IgE in serum.

## STATISTICAL METHODS:

A Statistical Analysis Plan (SAP) will be written prior to final database lock that will provide details on the planned statistical analysis. If discrepancies exist between the statistical analysis as described in the protocol and the final SAP, the SAP will prevail.

Safety and efficacy data will be merged and summarized with data from Study 190-201 to characterize the safety and efficacy of longer-term treatment. Safety assessments include adverse events, clinical laboratory results, vital signs, ECGs, and immunogenicity. Efficacy data include CLN2 assessments and MRI measurements of brain volumes.



190-202 Amendment 6

Page 10

# 3 TABLE OF CONTENTS

| 1 | TIT | LE PAG | E | 1 |
|---|---|---|---|---|
| 2 | SYN | NOPSIS. | | 4 |
| 3 | TABLE OF CONTENTS | | | 10 |
| 4 | ABBREVIATIONS | | | |
| 5 | | | | |
| | 5.1 | Institut | tional Review Board or Independent Ethics Committee | 16 |
| | 5.2 | | Conduct of Study | |
| | 5.3 | Subjec | t Information and Informed Consent | 17 |
| 6 | INV | _ | ATORS AND STUDY ADMINISTRATIVE STRUCTURE | |
| 7 | INT | RODUC | CTION | 20 |
| | 7.1 | Noncli | nical Studies | 20 |
| | 7.2 | Previo | us Clinical Studies | 21 |
| | 7.3 | Study 1 | Rationale | 23 |
| | 7.4 | Summa | ary of Overall Risks and Benefits | 24 |
| | | 7.4.1 | Hypersensitivity Reactions | 24 |
| | | 7.4.2 | Risks of Intracerebroventricular Devices and Drug Administration | 25 |
| 8 | STU | JDY OB | JECTIVES | 27 |
| 9 | INV | ESTIGA | ATIONAL PLAN | 28 |
| | 9.1 | Overal | l Study Design and Plan | 28 |
| | 9.2 Discussion of Study Design, Including Choice of Control Group | | 34 | |
| | 9.3 Selection of Study Population | | 34 | |
| | | 9.3.1 | Inclusion Criteria | 34 |
| | | 9.3.2 | Exclusion Criteria | 34 |
| | | 9.3.3 | Removal of Subjects from Treatment or Assessment | 35 |
| | | 9.3.4 | Subject Identification and Replacement of Subjects | 37 |
| | | 9.3.5 | Duration of Subject Participation | 37 |
| | 9.4 | Treatm | ents | 37 |
| | | 9.4.1 | Treatments Administered | 37 |
| | | 9.4.2 | Identity of Investigational Product | 38 |

| Bic | MP | ARIN | 190-202 Amendment 6 | Page 11 |
|---|---|---|---|---|
| | 9.4.3 | Storage | | 38 |
| | 9.4.4 | 9.4.4 Directions for Administration | | |
| | 9.4.5 | Method of | Method of Assigning Subjects to Treatment Groups | |
| | 9.4.6 | Selection of | Selection of Doses Used in the Study | |
| | 9.4.7 | Blinding | | 43 |
| | 9.4.8 | Prior and C | Prior and Concomitant Medications | |
| | 9.4.9 | Treatment | Compliance | 44 |
| 9.5 | Investig | gational Pro | duct Accountability | 44 |
| | 9.5.1 | Return and | Disposition of Clinical Supplies | 44 |
| 9.6 | Dietary | or Other Pr | rotocol Restrictions | 45 |
| 9.7 | Efficac | y and Safety | Variables | 45 |
| | 9.7.1 | Primary Et | ficacy Variables | 45 |
| | 9.7.2 | Secondary | Efficacy Variables | 46 |
| | 9.7.3 | Explorator | Exploratory Variables | |
| | 9.7.4 | Immunogenicity | | |
| | 9.7.5 | Safety Var | iables | 49 |
| | 9.7.6 | | s, Physical Examinations and Other Obs | |
| 10 REP | ORTING | G ADVERS | E EVENTS | 55 |
| 10.1 | Advers | e Events | | 55 |
| 10.2 | Serious | Adverse Ev | /ents | 59 |
| 10.3 | Advers | e Events of | Special Interest | 61 |
| 10.4 | Procedu | ares for Rec | ording Adverse Events | 61 |
| | 10.4.1 | Recording | Adverse Events on a eCRF | 61 |
| | 10.4.2 | Diagnosis | versus Signs and Symptoms | 62 |
| | 10.4.3 | Adverse E | vents Occurring Secondary to Other Eve | ents62 |
| | 10.4.4 | Persistent of | or Recurrent Adverse Events | 62 |
| | 10.4.5 | Abnormal | Laboratory Values | 62 |
| | 10.4.6 | Pre-existin | g Conditions | 63 |
| | 10.4.7 | General Ph | nysical Examination Findings | 63 |
| | 10.4.8 | Hospitaliza | ation, Prolonged Hospitalization, or Sur | gery64 |

| BEOMARIN | 190-202 Amendment 6 | Page 12 |
|---------------------------|--------------------------------|-----------|
| 10.4.9 Deaths | | 64 |
| 10.4.10 Pregnancy | | 64 |
| | Requirements | |
| 10.5 Urgent Safety Mea | sures | 65 |
| | ovigilance Contact Information | |
| 11 APPROPRIATENESS C | OF MEASUREMENTS | 67 |
| 11.1 Natural History Stu | ıdies | 67 |
| | ating Scales | |
| 11.3 Magnetic Resonance | ce Imaging | 68 |
| 12 STUDY PROCEDURES | S | 70 |
| 12.1 Screening/Baseline | · | 70 |
| 12.2 Treatment Visit(s). | | 70 |
| 12.2.1 Every Visi | t (every 2 weeks ± 3 days) | 70 |
| 12.2.2 Every 8 W | eeks | 71 |
| 12.2.3 Every 12 V | Weeks | 71 |
| 12.2.4 Every 24 V | Weeks | 72 |
| 12.2.5 Every 48 V | Veeks | 72 |
| 12.3 Study Completion | or Early Termination Visit | 72 |
| 12.4 Device Safety Follo | ow-Up | 73 |
| 12.5 Safety Follow-Up | | 74 |
| 12.6 Study Termination. | | 75 |
| 13 DATA QUALITY ASSU | JRANCE | 76 |
| 14 STATISTICAL METHO | DDS AND DETERMINATION OF SAMP | LE SIZE77 |
| 14.1 Statistical and Anal | lytical Plans | 77 |
| 14.1.1 Interim Ar | nalyses | 77 |
| 14.2 Primary Efficacy A | analysis | 77 |
| 14.3 Secondary Efficacy | / Analysis | 77 |
| 14.4 Exploratory Analys | ses | 77 |
| 14.5 Immunogenicity A | nalysis | 78 |
| 14.6 Safety Analysis | | 78 |

|---|---|---|
| 14.7 Determination of S | ample Size | |
| | nduct of the Study or Planned Analyses | |
| | COMMITTEE | |
| | SURANCE AND INDEMNITY | |
| | S AND SOURCE DOCUMENTS | |
| | G AND AUDITING | |
| | ORDS | |
| | ON AND PUBLICATION | |
| 21 REFERENCES | | 87 |
| | PONSIBILITIES | |
| | and Protection of Human Subjects | |
| 25 PROTOCOL AMENDM | MENT TEXT REVISIONS | 93 |
| | LIST OF TABLES | |
| Table 9.1.1: Schedule of Ev | ents | 30 |
| Table 9.7.5.3.1: Clinical La | boratory Tests | 51 |
| | Event Grading (Severity) Scale | |
| | Attribution Guidance | |
| | LIST OF APPENDICES | |
| Appendix 1: Adapted CLN | 2 Disease Rating Scale | 91 |



### 4 ABBREVIATIONS

AE adverse event

CBC complete blood count

CFR Code of Federal Regulations

CLN2 late-infantile neuronal ceroid lipofuscinosis disease, also known as classical late-infantile

CLN2, cLINCL, or Jansky-Bielschowsky disease, a form of Batten Disease

CNS central nervous system
CRA clinical research associate
CSF cerebrospinal fluid

CT computed tomography

CTCAE Common Terminology Criteria for Adverse Events

DBP diastolic blood pressure
DMC Data Monitoring Committee

ECG electrocardiogram

eCRF electronic case report form EEG electroencephalogram

ERT enzyme replacement therapy

EU European Union

EudraCT European Union Drug Regulating Authorities Clinical Trials

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB investigator brochure ICF informed consent form

ICH International Conference on Harmonisation of Technical Requirements for Registration of

Pharmaceuticals for Human Use

ICH E6 ICH Harmonised Tripartite Guideline: Guideline for Good Clinical Practice E6

ICV intracerebroventricular

IND Investigational New Drug (application)

IRB Institutional Review Board IEC Independent Ethics Committee

IP investigational product

MedDRA Medical Dictionary for Regulatory Activities

ML Combined score of motor and language subscales on the adapted CLN2 disease rating scale

MRI magnetic resonance imaging
MRS magnetic resonance spectroscopy
NAb neutralizing anti-TPP1 antibody

NCI National Cancer Institute

NOAEL no-observed-adverse-effect level OCT optical coherence tomography

PD pharmacodynamics



PedsQL measurement model for Pediatric Quality of Life Inventory

PICU pediatric intensive care unit

PK pharmacokinetics

PLT Preferential Looking Test

qow every other week
REB Research Ethics Board
SAE serious adverse event
SAR serious adverse reaction
SAP statistical analysis plan
SBP systolic blood pressure
SOC system organ class

SUSAR suspected unexpected serious adverse reaction

TAb total anti-TPP1 antibody TPP1 tripeptidyl peptidase 1

US United States

# **Definition of Terms:**

# Investigational Product (IP):

"A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use" (from International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use ICH Harmonised Tripartite Guideline: Guideline for Good Clinical Practice E6 [ICH E6]).

The terms "IP" and "study drug" may be used interchangeably in the protocol.

|----------|---------------------|---------|
|----------|---------------------|---------|

### 5 ETHICS

BioMarin Pharmaceutical Inc. (hereafter referred to as BioMarin or the Sponsor) conducts its studies according to the highest ethical and scientific standards. The following sections articulate standards to which Investigators will be held accountable, as well as matters of compliance to document adherence to such standards.

# 5.1 Institutional Review Board or Independent Ethics Committee

Investigators are expected to interact with Ethics Committees (ECs) promptly, as required, during the course of the study. This includes, but is not limited to, providing appropriate documentation to support study initiation and maintaining appropriate flow of safety and other information during the course of the study and for study close-out activities. BioMarin (or designee) will assist Investigators with access to timely and accurate information and with assurance of prompt resolution of any queries.

Prior to initiating the study, the Investigator will obtain written confirmation that the institutional review board (IRB), independent ethics committee (IEC), or Research Ethics Board (REB) (for Canadian protocols), is properly constituted and compliant with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) requirements, applicable laws and local regulations. A copy of the confirmation from the IRB/EC/REB will be provided to BioMarin Pharmaceutical Inc. (BioMarin) or its designee. The Investigator will provide the IRB/EC/REB with all appropriate material, including the protocol, Investigator's Brochure (IB), the Informed Consent Form (ICF) including compensation procedures, and any other written information provided to the subjects, including all ICFs translated to a language other than the native language of the clinical site. The study will not be initiated and Investigational Product (IP) supplies will not be shipped to the site until appropriate documents from the IRB/EC/REB confirming unconditional approval of the protocol, the ICF and all subject recruitment materials are obtained in writing by the Investigator and copies are received at BioMarin or its designee. The approval document should refer to the study by protocol title and BioMarin protocol number (if possible), identify the documents reviewed, and include the date of the review and approval. BioMarin will ensure that the appropriate reports on the progress of the study are made to the IRB/EC/REB and BioMarin by the Investigator in accordance with applicable guidance documents and governmental regulations.



# 5.2 Ethical Conduct of Study

It is expected that Investigators understand and comply with the protocol. This includes, but is not limited to: establishing and meeting enrollment commitments, including providing eligible subjects for study enrollment; adhering to diagnostic or other procedures as specified in the protocol; and assuring appropriate compliance with study treatment administration and accountability.

This study will be conducted in accordance with the following:

- US Code of Federal Regulations (CFR) sections that address clinical research studies, and/or other national and local regulations, as applicable
- Clinical Trial Directive 2001/20/EC and GCP Directive 2005/28/EC
- Other national and local regulations, as applicable
- ICH Harmonised Tripartite Guideline: Guideline for Good Clinical Practice E6 (ICH E6)
- The ethical principles established by the Declaration of Helsinki

Specifically, this study is based on adequately performed laboratory and animal experimentation. The study will be conducted under a protocol reviewed and approved by an IRB/EC/REB and will be conducted by scientifically and medically qualified persons. The benefits of the study are in proportion to the risks. The rights and welfare of the subjects will be respected and the investigators conducting the study do not find the hazards to outweigh the potential benefits. Each subject, or his/her legally authorized representative will provide written, informed consent before any study-related tests or evaluations are performed.

# 5.3 Subject Information and Informed Consent

A properly written and executed ICF, in compliance with the Declaration of Helsinki, ICH E6 (Section 4.8), United States (US) Code of Federal Regulations (CFR) 21 CFR §50, Directive 2001/20/EC, and other applicable local regulations, will be obtained for each subject prior to entering the subject into the study. The Investigator will prepare the ICF and provide the documents to BioMarin for approval prior to submission to the IRB/EC/REB approval. BioMarin and the IRB/EC/REB must approve the documents before they are implemented. A copy of the approved ICF (minor assent form and parental ICF for studies involving minors), and if applicable, a copy of the approved subject information sheet and all ICFs translated to a language other than the native language of the clinical site must also be received by BioMarin or designee prior to any study-specific procedures being performed.




Subjects under the age of 18 years will provide written assent (if required), and his/her legally authorized representative (parent or legal guardian) will provide written informed consent for such subjects. The Investigator will provide copies of the signed ICF to each subject (or the legally authorized representative of the subject) and will maintain the original in the record file of the subject.



## 6 INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

During administration of informed consent, expectations regarding participation in the study should be made clear to subjects. Subjects who are not willing and/or are not able to comply with all aspects of the study should not be encouraged to participate.

Prior to beginning the study, the Investigator at each site must provide to BioMarin or designee, a fully executed and signed US Food and Drug Administration (FDA) Form FDA 1572 and a Financial Disclosure Form. All sub-Investigators must be listed on Form FDA 1572. Financial Disclosure Forms must also be completed for all sub-Investigators listed on the Form FDA 1572 who will be directly involved in the treatment or evaluation of subjects in this study.

The study will be administered by and monitored by employees or representatives of BioMarin. Clinical Research Associates (CRAs) or trained designees will monitor each site on a periodic basis and perform verification of source documentation for each subject as well as other required review processes. BioMarin Pharmacovigilance (or designee) will be responsible for the timely reporting of serious adverse events (SAEs) to appropriate regulatory authorities as required.

In multicenter studies, a Coordinating Investigator will be identified who will be responsible for study overview. The Coordinating Investigator will read the clinical study report (CSR) and confirm that it accurately describes the conduct and results of the study, to the best of his or her knowledge. The Coordinating Investigator will be chosen on the basis of active participation in the study, ability to interpret data, and willingness to review and sign the report in a specified timeframe. The identity of the Coordinating Investigator and a list of all Investigators participating in the study will be provided in the CSR.

Assessment of immunogenicity and disease-related biomarkers will be conducted by BioMarin. Clinical laboratory evaluations will be performed by local study site laboratories. Central laboratories will be used to evaluate TPP1 enzyme activity, magnetic resonance imaging (MRI) scans, and electroencephalograms (EEGs). Additional details will be provided in the corresponding Study Laboratory Manual.



### 7 INTRODUCTION

CLN2 disease, also known as late-infantile neuronal ceroid lipofuscinosis, NCL type 2 or Jansky-Bielschowsky disease, is a form of Batten Disease, a group of rare fatal pediatric dementias. CLN2 is caused by the deficiency of TPP1, resulting from mutations in the *CLN2* gene. TPP1 functions in the cell lysosome to cleave N-terminal tripeptides from a number of substrates. In the absence of TPP1, materials normally metabolized by this enzyme form abnormal autofluorescent inclusions in cell lysosomes. The CNS is uniquely susceptible to this process and the disease manifests as a neurodegenerative disorder and, ultimately, death. The onset of clinical symptoms is typically between ages 2 and 4 (Chang, 2011); (Kurachi, 2000) with an average age of diagnosis of 4 years. Patients typically present initially with seizures, followed by ataxia, myoclonus, impaired speech, cognitive impairment, and developmental regression. A decline in vision and motor skills follows, with patients blind and wheelchair bound by approximately 6 to 8 years of age. Patients enter into a vegetative state during the later stages of the disease and feeding and tending to everyday needs become very difficult. Disease progression is very rapid with death typically occurring between 10 and 15 years of age.

## 7.1 Nonclinical Studies

Nonclinical studies indicate likely therapeutic benefit without significant risk of BMN 190-related toxicity for patients with CLN2 disease. In CLN2 disease animal models, after either intracerebroventricular (ICV) or intrathecal (via the cisterna magna and lumbar spine) administration, BMN 190 reduced lysosomal storage, attenuated functional decline, delayed disease progression, and extended lifespan. In TPP1 KO mice, restoration of TPP1 enzyme activity reduced lysosomal storage accumulation, improved motor function, and extended lifespan (Sleat, 2008); (Xu, 2011). In TPP1-null dachshunds, BMN 190 also reduced lysosomal storage, preserved function, and extended lifespan; in addition, onset of neurodegenerative clinical signs was delayed or prevented (Vuillemenot, 2011); (Katz, 2014) BMN 190-10-077). Studies in cynomolgus monkeys have indicated widespread distribution of active enzyme in the CNS after ICV infusion and no drug-related safety findings (Vuillemenot, 2014).

BMN 190 concentrations in cerebrospinal fluid (CSF) remained above the lysosomal K<sub>uptake</sub> for approximately 48 hours after single ICV or intrathecal infusions in species (dog and monkey) with CSF dynamics similar to those in human (Study BMN 190-09-071; Study BMN 190-10-077; Study BMN 190-11-046; Vuillemenot, 2014). In these same species, CNS distribution of BMN 190 was extensive in many brain regions. Distribution and PK



characteristics after ICV infusion of BMN 190 appear even more advantageous than intrathecal administration for treatment of CLN2 disease. A mean CNS half-life of approximately 2 weeks (range, 3.1 to 87.2 days, depending on CNS site) (BMN 190-09-071) suggests biweekly dosing may sustain therapeutic BMN 190 levels in the CNS.

Considered collectively, toxicology data have not identified any drug-related safety issues when BMN 190 is administered by ICV or intrathecal infusion to healthy animals or animals with CLN2 disease. Repeated BMN 190 administration was associated with inflammation and neuronal necrosis adjacent to the ventricles and ICV catheter track in dog (BMN 190-10-077) and was largely attributable to the implanted catheters and infusion procedure; vehicle-treated and wild-type treated animals exhibited the same findings. Hypersensitivity reactions in dachshunds following repeated BMN 190 administration, correlating with systemic exposure and anti-BMN 190 antibody titers, were attributed to the canine immune response to human heterologous protein and were clinically manageable with infusion time extension (BMN 190-10-077). Systemic toxicity due to exaggerated pharmacology is unlikely since BMN 190 is the inactive pro-form of human TPP1 that requires lysosomal uptake for activation. Also, the bulk of ICV-administered BMN 190 remains in the CNS.

Maximum ICV dose levels for monkey and dachshund studies were based on upper limits of BMN 190 concentration at the time of study initiation, infusion rate, and infusion time. Infusion conditions were selected to minimize effects on intracranial pressure due to rapid changes in CSF volume as well as to minimize the anesthetization period needed for the infusion procedure. Extension of the infusion time from 2 hours (at 0.6 mL/hour) to 4 hours (at 0.3 mL/hour) mitigated hypersensitivity reactions in dachshunds. An amount equivalent to approximately 5% of the total CSF volume was infused per hour in dog and monkey studies. Thus, the maximum feasible ICV doses were 16 mg/dose for dog (BMN 190-10-077) and 20 mg/dose for monkey (BMN 190-09-071).

### 7.2 Previous Clinical Studies

BMN 190 has been studied in human clinical trials 190-201 and 190-202. Study 190-201 was a 48-week, international, multicenter phase 1/2 open-label dose-escalation study designed to assess the safety and efficacy of BMN 190 administered to patients with mild to moderate CLN2 disease by direct intracerebroventricular infusion to the CNS; Study 190-202 is the open-label extension of 190-201.

These studies evaluated the safety, tolerability and efficacy of BMN 190 given as an infusion of 300 mg every 14 days given directly to the CNS using a permanently implanted



intracerebroventricular (ICV) access device. A total of 24 patients with screening CLN2 motor-language scores  $\geq 3$  (0 to 6 point scale) and age  $\geq 3$  were enrolled into the 190-201 study. All completers without predefined stopping criteria were qualified to enroll into the long term extension, Study 190-202.

All patients had successful surgical implantation of ICV access devices, with device complication rates consistent with what has been observed in the published literature.

Interim results of the completed 48-week open-label study (190-201) and the ongoing extension study (190-202) have been published (Schulz, 2018). The primary outcome measure was the time until a 2-point decline in the score on the motor and language domains of the CLN2 Clinical Rating Scale (which ranges from 0 to 6, with 0 representing no function and 3 representing normal function in each of the two domains), which was compared with the time until a 2-point decline in 42 historical controls. Additionally, rate of decline in motor—language score was compared between the two groups using data from baseline to the last assessment with a score of more than 0, divided by the length of follow-up (in units of 48 weeks).

Twenty-four subjects were enrolled in Study 190-201/ 190-202, 23 of whom constituted the efficacy population. Interim efficacy results demonstrated a statistically significant and durable treatment effect in attenuating disease progression as measured by CLN2 scores and in comparison to natural history. Of the 24 patients enrolled into Study190-201, all but 2 subjects were in the active loss of function phase of the disease characterized by both notable disease burden and decline by a median value of 2 points per 48 weeks. In the 23 subjects who received BMN 190 for at least 96 weeks in Study 190-201/ 190-202, the median time until a 2-point decline in the motor—language score was not reached and was 345 days for historical controls. The mean (SD) unadjusted rate of decline in the motor—language score per 48-week period was 0.27 (0.35) points in treated subjects and 2.12 (0.98) points in 42 historical controls (mean difference, 1.85; P < 0.001). Common AEs included convulsions, pyrexia, vomiting, hypersensitivity reactions, and failure of the intraventricular device. In 2 subjects, infections developed in the intraventricular device that was used to administer the infusion, which required antibiotic treatment and device replacement.

PK analysis of ICV-delivered BMN 190 demonstrates concentrations and exposures that are three orders of magnitude greater in the CSF than in the plasma.

No association was found between ADA, including drug-specific IgE positivity, and incidence or severity of hypersensitivity adverse events.



Taken together, the response in the treated group is significant when compared to the loss of function predicted by natural history studies. The conclusions of treatment effect are constant across all analysis methodologies and sensitivity analyses. Most patients (87%) experience neurodegenerative stabilization, in which active decline in function is either halted (57%), has an early single point decline with no subsequent loss (22%) or actually improves function on treatment (9%).

In conclusion, BMN 190 via ICV infusion is generally safe and well tolerated. BMN 190 treatment demonstrated a durable and clinically meaningful therapeutic effect on attenuating disease progression compared to natural history.

## 7.3 Study Rationale

BMN 190 is a recombinant form of human tripeptidyl peptidase 1(TPP1), the enzyme deficient in patients with CLN2 disease (also known as classical late-infantile CLN2, cLINCL, or Jansky-Bielschowsky disease), a form of Batten Disease. As an enzyme replacement therapy (ERT), BMN 190, is expected to restore TPP1 enzyme activity. Given the urgent and severe unmet medical need in CLN2 disease and observations in neurologically relevant animal models of CLN2 disease, clinical development of BMN 190 ERT is justified.

Murine and canine models of CLN2 disease (sharing the same genetic and enzymatic defect TPP1 deficiency, as the human disorder) recapitulate the major human clinical signs and pathology, including neuron loss, tremor, ataxia, functional decline, and reduced lifespan. (Awano, 2006); (Sleat, 2004). ERT with BMN 190 administered intrathecally in both models yielded pharmacologically significant benefit. Furthermore, when dosing started early in life (~2.5 months of age) in the TPP1-null dachshund model, BMN 190 significantly delayed onset of clinical signs, preserved motor and cognitive function, and prolonged life. The better pharmacological response to ERT in this and other animal models, when treatment was started closer to birth, indicates the importance of starting therapy as early in life as possible. (Dierenfeld, 2010).

There is currently no accepted, standard treatment for CLN2 other than supportive care. Enzyme replacement therapy (ERT) with BMN 190, or recombinant human TPP1 (rhTPP1), may be a potential new treatment option for CLN2 patients. BMN 190 is expected to reduce the progressive, pathologic accumulation of lysosomal storage material, and improve signs and symptoms of the disease.

The Phase 1/2 study (190-201) evaluated the efficacy and safety of doses up to 300 mg/every other week (qow) BMN 190 in patients with CLN2 disease. Results from the 190-201 study



demonstrated a substantial improvement of the rate of clinical progression in children treated with BMN 190 compared with untreated historical controls. Further, in those children who had received at least 48 weeks of BMN 190 dosing, clinical scores stabilized, in contrast to matched historical untreated controls in which decline was rapid and profound in the majority of matches.

The dose and regimen for this study (190-202) are based on the results of the 190-201 study. The rationale for this phase 2 extension study is to provide patients who complete the 190-201 study with the option to continue BMN 190 treatment. The 190-202 study is an open label extension protocol to assess long-term safety and efficacy.

## 7.4 Summary of Overall Risks and Benefits

Nonclinical toxicity studies have not identified drug-related adverse effects associated with chronic ICV administration of BMN 190 to healthy or CLN2 animal models disease.

BMN 190 has been studied in 24 patients in 5 clinical sites for Studies 190-201 and 190-202. The current clinical experience in human clinical trials demonstrates an acceptable benefit-risk profile to both the placement and chronic use of ICV access devices, and to infusion of BMN 190 at 300 mg every 14 days as demonstrated by interim efficacy and safety results summarized in Section 7.2. The efficacy objective of this study is to prevent patients from entering into the active rapid loss of function phase of the disease, or to attenuate further progression of disease. Monitoring and evaluation of specific adverse events of hypersensitivity reactions and device-related complications are discussed in Sections 7.4.1 and 7.4.2. Given the severity of disease, clinical and nonclinical support, the overall risks and benefits support this protocol.

## 7.4.1 Hypersensitivity Reactions

Hypersensitivity reactions, including anaphylaxis and less severe allergic reactions, are an identified risk for ERT in general, including BMN 190. Thus, anaphylaxis and less severe allergic reactions may occur during and following ICV infusion of BMN 190. Therefore, it is required that appropriately trained personnel and equipment for emergency resuscitation (including epinephrine) be available near the bedside during study drug infusion. For information regarding the reporting of hypersensitivity reactions, refer to Section 10.3.

An allergic reaction is a disorder characterized by an adverse local or general response from exposure to an allergen. Allergic reaction may include a combination of the following symptoms: flushing or rash, fever, urticaria, dyspnea, symptomatic bronchospasm with or without urticaria, allergy-related edema/angioedema, hypotension, or anaphylaxis. Infusion of BMN 190 may provoke additional symptoms of allergic reactions not included in this list.



The investigator will categorize the severity of an allergic reaction as described in Section 10.1.

Anaphylaxis, a systemic, immediate hypersensitivity reaction, is the most severe form of hypersensitivity reaction. Symptoms may occur during or within hours following infusion of an agent and, generally, more rapid onset indicates more severe reaction; death may result. Managing anaphylaxis requires early recognition of signs and symptoms and clinicians well trained in the management of acute events. Symptoms of anaphylaxis may include involvement of skin and/or mucosal tissue (e.g., generalized hives, pruritus or flushing, swollen lips-tongue-uvula) respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia), and reduced blood pressure or end-organ dysfunction (e.g., hypotonia, syncope, incontinence).

All AEs, including hypersensitivity, anaphylaxis and other allergic reactions that occur within 24 hours after infusion start or restart, regardless of the investigator's assessment of study drug relationship, will be assessed to be hypersensitivity reactions. It is expected that the adverse events of greatest clinical importance will be immune-mediated hypersensitivity reactions, but not all hypersensitivity reactions may be allergic in nature. The risk of such reactions may be mitigated by specific measures, including pretreatment or infusion modification, as described in Section 9.4.4.

# 7.4.2 Risks of Intracerebroventricular Devices and Drug Administration

Patients in this study will have had an ICV reservoir surgically implanted for administration of BMN 190. The use of ICV devices may result in infections, intracerebral hemorrhage reservoir leakage, and seizures (Karavelis, 1996), (Kronenberg, 1998). Additional surgery may be required to fix or replace the devices. The technical complication rate of one ICV reservoir study in 106 cancer patients was 10.3% with almost half of these complications requiring surgical revision (median time reservoirs were in place was 4.1 months ranging from 2 days to 4.6 years) (Lishner, 1990). Although these devices have been approved for use for decades, there is little available safety data for long term use.

Patients will be monitored throughout the study for potential infections (high temperature, cough, rash, headache, mental status changes, swelling or drainage in the incision area) and signs of ICV reservoir leakage or failure (swelling of skin around reservoir site, difficulty with CSF extraction, erythema of the scalp, bulging of reservoir device, or extravasation of fluid on infusion).

The investigator will evaluate the patency, location, and skin integrity of the reservoir at each study drug administration. The investigator will check for scalp edema, erythema or skin



breakdown at the site of the reservoir prior to infusion. Patency will be assessed during pre-infusion sampling and again at the time of infusion. Difficulty in obtaining the required volume of CSF needed for pre-infusion samples or signs of ICV reservoir leakage (swelling of skin around reservoir site, erythema of the scalp, bulging of reservoir device, or extravasation of fluid) will prompt further evaluation of the reservoir for failure prior to continuing with infusion. Additional surgical consultation including surgery may be required to fix or replace the device (refer to Section 9.7.6.2). Material degradation of the ICV device reservoir has occurred after approximately 105 perforations of the ICV device in benchtop testing, and has been observed in clinical trials with approximately 4 years of BMN 190 administration. Access device replacement should be considered prior to 4 years of regular administration of BMN 190; with the decision made on an individual subject level based on the medical judgment of the Investigator.

All BMN 190 infusions are given in an inpatient setting with supportive measures present. A follow-up phone call will be conducted ~48 hours after the patient has been discharged from each infusion visit.

|----------|---------------------|---------|
|----------|---------------------|---------|

### 8 STUDY OBJECTIVES

The primary objective of the study is:

- To evaluate the long-term safety of BMN 190 administration at 300 mg qow in patients with CLN2.
- To assess change in motor and language (ML) subscales of the CLN2 disease rating scale in patients with CLN2 receiving BMN 190 at 300 mg qow.

The secondary objectives of the study are:

- To assess changes in quantitative assessment of MRI.
- To assess change in CLN2 disease scale total score.
- To evaluate quality of life (QoL) with long-term BMN 190 administration.

The exploratory objectives of the study are:

- To evaluate age-appropriate developmental milestones with long-term BMN 190 administration.
- To evaluate the impact of treatment on disease-related biomarkers from CSF and blood.



### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

This is a multi-center, multinational, extension study to evaluate BMN 190 treatment in patients with CLN2 who completed 190-201. All patients who have completed 48 weeks in Study 190-201 will be eligible to enroll in Study 190-202.

The Screening period for Study 190-202 will start simultaneously with the Week 47 visit in Study 190-201. Baseline values for Study 190-202 will be recorded at the first infusion, Week 1 Day 1 of Study BMN 190-202, for all patients on active treatment. The first dose of BMN 190 in Study 190-202 (Week 1/Study Day 1) will be given following the Week 49 study assessments in Study 190-201. This study will be open label with all patients continuing on treatment with BMN 190 300 mg qow.

Patients will complete safety and efficacy assessments including CSF surveillance labs every 2 weeks, CLN2 disease scales every 8 weeks, clinical laboratory assessments, visual acuity tests, and immunogenicity tests every 12 weeks. MRI, quality of life measures, OCT, EEG, developmental milestones (Denver II), and blood and CSF samples for evaluating disease-related biomarkers will be collected every 24 weeks. Complete physical examination will be performed every 48 weeks.

Some patients may experience hypersensitivity reactions associated with the administration of study drug, thus prophylactic antihistamine may be administered prior to each study drug infusion at the discretion of the Investigator. Antipyretic pretreatment may be given at the Investigator's discretion. Vital signs will be measured just before, during, and immediately following the study-drug infusion. Adverse events and changes in concomitant medication will be recorded throughout the study.

To date there has been no anaphylaxis or anaphylactoid reactions in studies with BMN 190. However, in the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion).

In addition, the investigator must contact the BioMarin medical monitor (Section 10.6) within 1 business day if any AE is severe (Grade 3 or higher) or serious <u>and</u> requires any of the following:

• infusion interruption, discontinuation, or modification (not due to blocked line)



- administration of IV fluids, steroids, or antihistamines
- administration of oxygen

Before subsequent infusions, the investigator and BioMarin medical monitor will discuss the case and agree upon infusion modification or additional premedication. Agreed upon dose modifications or introduction of additional premedication should be documented in the Electronic Case Report Forms (eCRFs) and source files.

Patients may withdraw voluntarily from receiving study drug at any time, and they may also withdraw entirely from complete study participation at any time, upon request. If BMN 190 treatment is suspended, BMN 190 may resume if no more than 2 consecutive doses are missed after the last given dose.

A summary of events and assessments are provided by visit in Table 9.1.1.



**Table 9.1.1: Schedule of Events** 

| Assessments and Events | Screening<br>Period<br>(2 weeks) | Q2<br>Weeks<br>± 3 days | Q8<br>Weeks | Q12<br>Weeks | Q24<br>Weeks | Q48<br>Weeks<br>± 3 days | Study Completion or ETV (2 weeks) ± 3 days after Week 239 | Device Safety Follow-Up (4 weeks after device removal) ± 3 days | Safety Follow-Up<br>(6 months after<br>last dose) |
|---|---|---|---|---|---|---|---|---|---|
| Informed consent/assent <sup>a</sup> | X | ± 3 days | ± 3 days | ± 3 days | ± 3 days | | WEEK 239 | ± 3 days | ±1 week |
| Criteria for study entry <sup>b</sup> | X | | | | | | | | |
| Medical history <sup>c</sup> | | X<br>(Week<br>1 only) | | | | | | | |
| CLN2 disease rating scales <sup>d</sup> | | | X | | | | X | X | X |
| Videotaping of CLN2 scales <sup>d</sup> | | | | | X | | X | | |
| Visual acuity testing <sup>e</sup> | | | | X | | | X | | |
| Optical coherence tomography <sup>f</sup> | | | | | X | | X | | |
| ECG (3- or 5-lead) <sup>g</sup> | | Xg | | | | | | | |
| ECG (12-lead) <sup>h</sup> | | X | | | X | | X | | X |
| EEG, standard awake <sup>i</sup> | | | | | X | | X | | X |
| MRI <sup>j</sup> | | | | | X | | X | | |
| CSF (cell count, protein, glucose, culture) <sup>k</sup> | | X | | | | | X | | |
| Device Patency/Infection <sup>1</sup> | | X | | | | | | | |
| Administer study drug | | X | | | | | | | |
| Phone follow-up <sup>m</sup> | | X | | | | | | | |
| CSF/blood for disease-related biomarkers <sup>n</sup> | | | | | X | | X | | |
| CSF/serum for immunogenicity <sup>o</sup> | | | | X | | | X | X | X |



| | Screening | Q2<br>Weeks | Q8<br>Weeks | Q12<br>Weeks | Q24<br>Weeks | Q48<br>Weeks | Study<br>Completion or<br>ETV<br>(2 weeks) | Device Safety<br>Follow-Up<br>(4 weeks after<br>device removal) | Safety Follow-Up<br>(6 months after<br>last dose) |
|---|---|---|---|---|---|---|---|---|---|
| Assessments and Events | Period (2 weeks) | ± 3 days | ± 3 days | ± 3 days | ± 3 days | ± 3 days | ± 3 days after<br>Week 239 | ± 3 days | ±1 week |
| | | | | | | | | (serum only) | (serum only) |
| Vital signs <sup>p</sup> | | X | | | | | X | X | X |
| Height/weight | | | | | X | | X | | X |
| Complete physical examination <sup>q</sup> | | | | | | X | X | | X |
| Brief physical examination <sup>r</sup> | | X | | | | | | X | |
| Blood/urine for clinical lab tests <sup>s</sup> | | | | X | | | X | X | X |
| CLN2 specific QoL questionnaire <sup>t</sup> | | | | | X | | X | | |
| PedsQL <sup>t</sup> | | | | | X | | X | | |
| Denver II Developmental Scale <sup>u</sup> | | | | | X | | X | | |
| Neurological examination | | | | X | | | X | X | |
| Pregnancy testing (in females of childbearing potential) <sup>v</sup> | X | | | | | | | | |
| Adverse events <sup>w</sup> | X | X | | | | | X | X | X |
| Concomitant medications | X | X | | | | | X | X | X |
| Hypersensitivity labs | | X <sup>x</sup> | | | | | | | |
| ICV Access device removal | | | | | | | X <sup>y</sup> | | |

Baseline values will be recorded at the time of the first infusion, Week 1 Day 1 of Study BMN 190-202. Thereafter, study visits will be every two weeks ±3 days. If done on the same day, assessments of function and QoL should precede MRI and blood and CSF sampling, which should precede infusion; sample collection may occur when subjects are sedated for MRI. If a subject is discontinued from the study prematurely, an Early Termination visit should be scheduled within 7 days.

<sup>&</sup>lt;sup>a</sup> Written informed consent must be obtained before study procedures begin.

<sup>&</sup>lt;sup>b</sup> Two domains (motor and language) of the Hamburg Scale will be tested for eligibility to enroll in 190-202. Subjects must not have had a loss of 3 or more points in the combined motor and language components at the end of 190-201 compared with 190-201 Baseline, and they also must not have a score of 0 on the combined motor and language components of the CLN2 rating scale.

|----------|---------------------|---------|
|----------|---------------------|---------|

- <sup>c</sup> Medical History to be collected during Week 1 only, and prior to receiving the first dose on 190-202. Any ongoing AEs/SAEs in 190-201 will be documented as medical history in 190-202.
- d All domains of both Hamburg Scale and Weill Cornell Scale will be tested every 8 weeks during the study through study completion (or within one week of Early Termination visit), at the 4-week Device Safety follow-up, and at the 6-month Safety follow-up visit. If done on the same day, assessments of function and QoL should precede MRI and blood and CSF sampling. Videotaping of the CLN2 disease scale evaluation will occur every 24 weeks when the CLN2 disease scale is assessed, at any time a Termination from the study is warranted, and at the first visit for all new sites.
- e All subjects will undergo Preferential Looking Testing every 12 weeks. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or E Hook (or Tumbling E) Vision Test should also be performed during the same assessment. Visual acuity testing can be performed either before or after the infusion (± 3 days), but should be performed at a time (relative to infusion) that can be repeated consistently between study visits. The subject must not be sedated at the time of visual acuity testing.
- f OCT should precede infusions. In order to limit the need for sedation to perform this assessment, measurement should be obtained while the subject is also under sedation for MRI acquisition.
- g For at least one infusion of BMN 190 (and preferably the next infusion), continuous ECG monitoring (3- or 5-lead) will be performed for all subjects. The ECG should begin 15 (± 5 minutes) prior to infusion start, continue through infusion of BMN 190, and end after infusion of flushing solution. If a 12-lead ECG is required during this time, continuous monitoring should be interrupted in order to obtain the 12-lead ECG.
- h A standard ECG (12-lead), including heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities, will be performed 30 (±5) minutes after infusion end at the first infusion and every 24 weeks thereafter. In patients with present or past bradycardia, conduction disorders, or with structural heart disease, an ECG will be performed within 30 minutes before the start of infusion (±5 minutes), at 2 hours (±15 minutes) during infusion, 30 (±5) minutes after infusion end, and 12 hours (±3 hours) after infusion end for each study drug infusion.
- <sup>i</sup> EEG values will be recorded within 2 days before each infusion at the specified time points.
- <sup>j</sup>MRI assessment should precede blood and CSF sampling. A ±4-week window is allowed for this assessment and may be performed at the same time as a scheduled infusion.
- <sup>k</sup> CSF (for cell count with differential, protein, glucose, and culture) will be collected within 30 (±5) minutes before every infusion (or within one week of the Early Termination visit).
- <sup>1</sup>Device and surgical location of the device should be observed prior to each infusion for any swelling or signs of infection of the scalp or surrounding area.
- m Parent/guardian will be telephoned ~48 hours for follow-up after having been discharged from each visit to document health status and to remind them to initiate contact if any symptom of concern is observed. At a minimum, the telephone follow up will include guidance for the parent or legal guardian to detect clinical signs of an infection of the ICV reservoir and meningitis or encephalitis.
- <sup>n</sup> Samples of blood and CSF will be collected prior to infusion.
- o Samples of blood (serum) and CSF will be collected for TAb and NAb testing before the first infusion (Study 190-201 Study Completion Visit), every 12 weeks thereafter, and at the Study Completion Visit of Study 190-202. Samples of blood (serum) will be collected for TAb testing at the Device Safety Follow-Up and Safety Follow-Up visits (or within 1 week of the Early Termination visit). Collection must precede infusion. Serum and CSF NAb will be tested prior to the first infusion (Study 190-201 Study Completion Visit) and at subsequent time points when serum and CSF TAb are positive, respectively. Samples from the Study Completion visit in Study 190-201 will be used to obtain a baseline

|----------|---------------------|---------|
|----------|---------------------|---------|

total and drug-specific IgE levels in the event of later hypersensitivity reactions requiring additional lab work. Samples of blood (serum) only will be collected for TAb, total IgE, C4, and tryptase as part of the Safety Follow-Up visit and the Device Safety Follow-Up visit; CSF will not be collected at either of these safety follow-up visits.

- P Vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], heart rate, respiration rate, and temperature) will be measured within 30 (±5) minutes before infusion start (or restart), every 30 (±5) minutes during infusion, 0.5 hours (±5 minutes), 1 hour (±5 minutes), and 4 hours (±15 minutes) after infusion end, and then every 4 hours (±15 minutes) for the next 16 hours. Blood pressure will be measured in the upper arm using an appropriately sized blood pressure cuff. If the patient's blood pressure is abnormal (as compared to site-specific reference ranges), a manual blood pressure will be obtained by a trained healthcare professional.
- <sup>q</sup> A <u>complete</u> physical examination will include general appearance, cardiovascular, dermatologic, lymphatic, respiratory, gastrointestinal, genitourinary, musculoskeletal, and neurologic systems. Clinically significant abnormalities will be recorded as AEs.
- <sup>r</sup> A <u>brief</u> physical examination will include general appearance, cardiovascular, respiratory, neurologic, and gastrointestinal systems. Clinically significant abnormalities will be recorded as AEs.
- <sup>s</sup> Samples for clinical laboratory assessments (hematology, chemistry, and urinalysis) will be collected before infusion.
- <sup>t</sup> Quality of life assessments include the PedsQL (including both a Parent Report for Toddlers and a Family Impact Module) and a CLN2 disease-based QoL instrument. If done on the same day, assessment of QoL should precede MRI and sampling.
- <sup>u</sup> If done the same day, assessment of function on the Denver II Developmental Scale should precede MRI and sampling.
- <sup>v</sup> During the Screening period, a female subject judged by the investigator to be of childbearing potential will be tested for pregnancy with a urine pregnancy test; additional urine tests will be performed during the study whenever pregnancy is in question. A serum pregnancy test will be performed if a urine test result is positive or equivocal.
- We All AEs and SAEs will be recorded starting with the first dose of study drug in Study 190-202 until 6 months after either the last administration of study drug or the Early Termination visit. A Safety Follow-Up visit will also be performed within 6 months after the last administration of study drug or Early Termination. The 6-month Safety Follow-Up Visit will be waived for subjects who begin receiving study drug in another BioMarin-sponsored study or registry within this 6-month period. Refer to Section 10.1 for AE and Section 10.2 for SAE reporting instructions for subjects who receive study drug in another BioMarin-sponsored study or registry within the 6-month period. For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week Device Safety and 6-month Safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug.
- <sup>x</sup> In the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion).
- y Following either the study completion visit (Week 239) or the Early Termination Visit, arrangements should be made for removal of the ICV access device. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, should also be returned. If the subject intends to continue to receive BMN 190 following participation in this study (e.g., via commercial product, use in a registry, or another BMN 190 study), then the device does not need to be removed. Device removal should occur no more than 4 weeks after the last administration of study drug. A device removal safety follow-up visit will be performed within 4 weeks (±3 days) from removal of the ICV access device.



# 9.2 Discussion of Study Design, Including Choice of Control Group

Study 190-202 is designed to be an extension for patients who complete 48 weeks in Study 190-201. Natural history data as collected in Study 190-901 will be used as a control group for comparison.

# 9.3 Selection of Study Population

All patients who have completed 48 weeks in Study 190-201 will be eligible to enroll in Study 190-202.

### 9.3.1 Inclusion Criteria

Individuals eligible to participate in this study must meet all of the following criteria:

- Must have completed 48 weeks in Study 190-201.
- Is willing and able to provide written, signed informed consent. Or, in the case of patients under the age of 18 (or other age as defined by regional law or regulation), provide written assent (if required) and have written informed consent, signed by a legally authorized representative, after the nature of the study has been explained, and prior to performance of research-related procedures.
- Males and females who are of reproductive age should practice true abstinence, defined as no sexual activity, during the study and for 6 months after the study has been completed (or withdrawal from the study). If sexually active and not practicing true abstinence, males and females of reproductive age must use a highly effective method of contraception while participating in the study.
- If female, of childbearing potential, must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests done during the study.

## 9.3.2 Exclusion Criteria

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

- Has had a loss of 3 or more points in the combined motor and language components of the Hamburg CLN2 rating scale between Baseline of Study 190-201 and the Study Completion visit in Study 190-201 and would not benefit from enrolling in the study in the Investigator's discretion.
- Has a score of 0 points on the combined motor and language components of the Hamburg CLN2 rating scale.
- Is pregnant or breastfeeding, at Baseline, or planning to become pregnant (self or partner) at any time during the study.



- Has used any investigational product (other than BMN 190 in 190-201), or investigational medical device, within 30 days prior to Baseline; or is required to use any investigational agent prior to completion of all scheduled study assessments.
- Has a concurrent disease or condition that would interfere with study participation, or pose a safety risk, as determined by the Investigator.
- Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

# 9.3.3 Removal of Subjects from Treatment or Assessment

Subjects (or their legally authorized representatives) may withdraw consent for study participation any time without prejudice; investigators must withdraw from the study any such subject. At the discretion of investigator clinical judgment, a subject may be withdrawn from the study any time. When possible, an Early Termination visit (ETV) should be completed (Section 12.6).

The investigator (or designee) must contact the BioMarin medical monitor when a subject discontinues from the study. BioMarin reserves the right to discontinue the study at any time for either clinical or administrative reasons and to discontinue participation of an individual investigator or study site for poor enrollment or noncompliance with the protocol or regulatory requirements. Subjects who discontinue from the study will have their reservoir and any associated hardware removed, unless doing so would be more harmful than not in the opinion of the Investigator or neurosurgeon.

Reasons for which the investigator or BioMarin may withdraw a subject from the study include, but are not limited to, the following:

- Subject experiences a serious or intolerable AE
- Subject develops a clinically significant laboratory abnormality
- Subject requires medication or medical procedure prohibited by the protocol
- Subject does not adhere to study requirements specified in the protocol
- Subject was erroneously admitted into the study or does not meet entry criteria
- Subject is lost to follow-up

If a subject fails to return for a scheduled visit, a documented effort must be made to determine the reason. If the subject cannot be reached by telephone, a certified letter should be sent to the subject (or the subject's legally authorized representative, if appropriate) requesting that s/he contact the investigator. A copy of this letter and any response should be


kept in the study records. If the subject cannot be contacted or fails to respond, the subject will be considered lost to follow-up.

The investigator (or designee) must explain to each subject before enrollment in the study that the subject's protected health information obtained during the study may be shared with the study sponsor, regulatory agencies, and IRB/IEC/REB. It is the responsibility of the investigator (or designee) to obtain written permission to use protected health information per country-specific regulations, such as HIPAA in the US, from each subject or (legally authorized representative, if appropriate). If permission to use protected health information is withdrawn, it is the investigator's responsibility to obtain a written request to ensure that no further data will be collected from the subject, and the subject will be removed from the study.

### 9.3.3.1 Stopping Criteria

As described in Section 10.1, all AEs, including toxicity of study drug, will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse AEs (CTCAE) v. 4.0.

Hypersensitivity reactions, including anaphylaxis and less severe allergic reactions, are identified risks of ERT. For hypersensitivity or allergic-type reactions, unacceptable drug-related toxicity shall be defined as a NCI CTCAE v. 4.0 Grade 3 or higher AE that is study-drug related in the opinion of the investigator and meets either of the following criteria:

- Shows no improvement with medical intervention, such as infusion interruption, infusion rate reduction, or administration of intravenous antihistamine, oxygen, intravenous fluids, or steroids; or
- Recurs during subsequent infusions at the same or worse severity and intensity, despite any of the following: premedication with appropriate antihistamines, antipyretics, or steroids; and modification of infusion rate.

Instances of unacceptable drug-related toxicity should be discussed by the investigator with the BioMarin medical monitor. A subject who experiences unacceptable drug-related toxicity may be withdrawn from study treatment after consultation with the BioMarin medical monitor.

Subjects who have a loss of 3 or more points on the combined motor and language components of the Hamburg CLN2 rating scale in any 1 year period may be discontinued at the discretion of the Investigator.



Subjects with a score of 0 on the combined motor and language components of the Hamburg CLN2 rating scale at two consecutive visits will be discontinued from treatment.

## 9.3.4 Subject Identification and Replacement of Subjects

Each subject will be assigned the same patient identifier that was used in Study 190-201, which will be on all eCRF pages. If the subject transfers primary study site between Study 190-201 and Study 190-202, the site number in the subject ID (first four numbers) will be updated, but the subject number (last four numbers) will remain the same. In legal jurisdictions where use of initials is not permitted, a substitute identifier will be used. Subjects who discontinue from the study for any reason will not be replaced.

#### 9.3.5 Duration of Subject Participation

Patients will receive qow ICV infusions of study drug, up to Week 239 or until one of the following occurs: the patient withdraws consent and discontinues from the study; the patient is discontinued from the study at the discretion of the Investigator; or the study is terminated in the region where the patient is being followed.

A Safety Follow-Up visit will be conducted 6 months after the final BMN 190 infusion. The Safety Follow-Up visit will be waived for subjects who receive study drug in another BioMarin-sponsored study or registry within this 6-month period (refer to Section 10.1 and Section 10.2 for AE and SAE reporting instructions). For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug.

#### 9.4 Treatments

BioMarin or its designee will provide the study site with study drug sufficient for study completion. BioMarin or its designee is responsible for shipping study drug to clinical sites.

#### 9.4.1 Treatments Administered

All study subjects will be administered BMN 190 300 mg by ICV infusion every two weeks (preferably in the morning). Fasting for a minimum of 2 hours before each infusion may be considered until the subject's reaction to the study drug is determined. When a feeding tube is used for an overnight feed, the tube may be turned off 2 hours before infusion.



## 9.4.2 Identity of Investigational Product

## 9.4.2.1 Product Characteristics and Labeling

The study drug label includes the following information: lot number, required storage conditions, a precautionary statement, expiry date, study number, and BioMarin name and address.

#### **9.4.3 Storage**

At the study site, all study drug must be stored under conditions specified in the Investigator's Brochure and BioMarin provided Pharmacy Manual in a secure area accessible only to the designated pharmacists and clinical site personnel. All study drug must be stored and inventoried, and inventories must be carefully and accurately documented according to applicable local, state, and federal regulations, ICH GCP, and study procedures.

#### 9.4.4 Directions for Administration

All study subjects will be administered BMN 190 300 mg by ICV infusion every two weeks (preferably in the morning). Fasting for a minimum of 2 hours before each infusion may be considered until the subject's reaction to the study drug is determined. When a feeding tube is used for an overnight feed, the tube may be turned off 2 hours before infusion. Study procedures for each study visit should precede study drug infusion unless otherwise specified. The date, time, volume, and concentration of each dose of study drug administered to each subject will be recorded in the dispensing log provided for the study as well as on the appropriate eCRF. The Study Pharmacy Manual provides further instructions on preparation and administration of study drug.

Subjects will be admitted to the hospital for every BMN 190 infusion. Subjects should be closely monitored in an appropriate inpatient setting for up to 48 hours following the start of each infusion; if no safety issues are observed, a subject may be discharged 24 hours after the infusion begins. Because hypersensitivity reactions may be associated with ERT administration, subjects may be pretreated with age-appropriate doses of antihistamine (and antipyretic, if appropriate) medication approximately 30 minutes (± 15 minutes) before BMN 190 infusion at the discretion of the investigator. Subjects may be pretreated, at the discretion of the Investigator, with age-appropriate sedative medication approximately 30 minutes (± 15 minutes) before BMN 190 infusion according to institution's standard practices. Clinical, developmental, and QoL assessments are to be performed before infusions.



BMN 190 will be infused ICV at 2.5 mL/hour to deliver the entire volume over approximately 4 hours. Uniform infusion rate should be ensured by use of a syringe pump with appropriate delivery range, delivery rate accuracy, and alarms for incorrect delivery or occlusion. If the dose needs to be stopped for safety or other reasons, it may be restarted at the same rate and completed so long as the total dose is administered within 10 hours of preparation.

At each administration, the investigator will draw 1-2 ml of CSF into the device cannula to check for patency prior to administering the study drug. This volume of CSF is also to be used for laboratory testing (cell count, protein, glucose, and culture) as noted in Table 9.1.1. Access to the device is performed using strict sterile technique. Skin covering the reservoir is inspected for an appropriate needle insertion site. The needle insertion site must be intact, without evidence of breakdown, wound, infection or rash. The needle used is a small gauge non-boring tip. Once the reservoir has been accessed, the needle is immobilized to ensure minimal movement or risk of removal. If the needle dislodges during an infusion, it may not be reinserted, as sterility has been compromised. At the discretion of the investigator and/or neurosurgeon, the reservoir may be replaced during the clinical study. Refer to Section 7.4.2 for risks associated with the implantation procedure.

All study subjects will be administered BMN 190 300 mg every other week. Doses lower than 300 mg may be administered at the discretion of the Investigator and upon consultation with the Medical Monitor if required for safety or other reasons.

#### 9.4.4.1 Safety Monitoring

Subjects will be admitted to the hospital for every BMN 190 infusion. For all infusions, subjects will be monitored in an appropriate inpatient setting for a minimum of 24 hours from the start of the infusion. A follow-up telephone call will be conducted ~48 hours after the subject has been discharged from the visit.

Vital signs (Section 9.7.6.1) will be measured at least at the following time points: within  $30 \ (\pm 5)$  minutes before infusion start (or restart), every  $30 \ (\pm 5)$  minutes during infusion, 0.5 hours ( $\pm 5$  minutes), 1 hour ( $\pm 5$  minutes), and 4 hours ( $\pm 15$  minutes) after infusion end, and then every 4 hours ( $\pm 15$  minutes) for the next 16 hours. Blood pressure will be measured in the upper arm using an appropriately sized blood pressure cuff. If the patient's blood pressure is abnormal (as compared to site-specific reference ranges), a manual blood pressure will be obtained by a trained healthcare professional.



For at least one infusion of BMN 190 (and preferably the next infusion), continuous ECG monitoring (3- or 5-lead) will be performed for all subjects. The ECG should begin 15 (±5 minutes) prior to infusion start, continue through infusion of BMN 190, and end after infusion of flushing solution. If a 12-lead ECG is required during this time, continuous monitoring should be interrupted in order to obtain the 12-lead ECG.

A standard ECG (12-lead), including heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities, will be performed 30 (±5) minutes after infusion end at the first infusion and every 24 weeks thereafter (Table 9.1.1). In patients with present or past bradycardia, conduction disorders, or with structural heart disease, an ECG will be performed within 30 minutes before the start of infusion (±5 minutes), at 2 hours (±15 minutes) during infusion, 30 (±5) minutes after infusion end, and 12 hours (±3 hours) after infusion end for each study drug infusion.

Subjects require regular monitoring for adverse events and epileptic seizures by appropriately trained personnel throughout the duration of the infusion. If epileptic seizures or any adverse events develop, the infusion may be interrupted at the discretion of the investigator. Because hypersensitivity reactions (anaphylaxis or general allergic) may occur, it is required that appropriately trained personnel and equipment for emergency resuscitation (including epinephrine) be available near the bedside during study drug infusion. In case emergency treatment is needed, all subjects should have an intravenous line during infusion. If the prior 3 study drug infusions were completed without significant adverse events, an intravenous access line does not have to be placed prior to infusion as consistent with local hospital policies. However, supplies for placing emergency access and all emergency medication must be readily available should they be needed. For information regarding the reporting of hypersensitivity reactions including anaphylaxis and other allergic reactions, refer to Section 10.3.

Symptoms of hypersensitivity reactions including anaphylaxis and other allergic reactions may include fever, chills/rigors, skin symptoms (urticaria, angioedema, rash), respiratory symptoms (dyspnea, wheezing, stridor), gastrointestinal symptoms (nausea, vomiting, abdominal pain), and/or cardiovascular changes (hypotension/hypertension). If more severe symptoms, such as angioedema (tongue or throat swelling) or stridor, develop, the infusion should be stopped.

To date, there has been no anaphylaxis or anaphylactoid reactions in studies with BMN 190. However, in the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood



samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion). Based on previous hypersensitivity reactions, and with the approval of the medical monitor, additional blood samples may be required following subsequent hypersensitivity reactions. Safety assessments will be conducted during and after each infusion. Subjects may be required to stay for a longer observation period at the investigator's discretion. If an AE consistent with a hypersensitivity reaction (Section 7.3) is observed, appropriate intervention may include infusion interruption, infusion rate decrease, or administration of antihistamine, oxygen, fluids, or steroids. If infusion is restarted after interruption, the initial rate should be approximately one-half the rate at which the hypersensitivity reaction occurred. Further detail for infusion modification is provided in the Study Pharmacy Manual.

The parent or legal guardian will be instructed to contact the investigator to discuss any AE subsequent to discharge.

The use of ICV devices can result in infections, intracerebral hemorrhage from chronic reservoir use, reservoir leakage, and seizures (Karavelis, 1996), (Kronenberg, 1998). Additional surgery may be required to fix or replace the devices. Patients will be monitored throughout the study for potential infections (high temperature, cough, rash, headache, swelling or drainage in the incision area) and signs of ICV reservoir leakage or failure (swelling of skin around reservoir site, difficulty with CSF extraction, erythema of the scalp, bulging of reservoir device, or extravasation of fluid on infusion).

The investigator will evaluate the patency, location, and skin integrity of the reservoir at each study drug administration. The investigator will check for scalp edema, erythema or skin breakdown at the site of the reservoir prior to infusion. Patency will be assessed during pre-infusion sampling and again at the time of infusion. Difficulty in obtaining the required volume of CSF needed for pre-infusion samples or signs of ICV reservoir leakage (swelling of skin around reservoir site, erythema of the scalp, bulging of reservoir device, or extravasation of fluid) will prompt further evaluation of the reservoir for failure prior to continuing with infusion. Additional surgical consultation including surgery may be required to fix or replace the device. In the event that the device is replaced, the next drug infusion will occur at least 14 days and no more than 28 days from surgery. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, should also be returned.



Because of the inherent safety considerations surrounding the implanted device, arrangements should be made for the subject to have the ICV access device removed no more than 4 weeks after either the Study Completion visit or the Early Termination visit. If the subject intends to continue to receive BMN 190 following participation in this study (eg., via commercial product, use in a registry, or another BMN 190 study), then the device does not need to be removed. A device removal safety follow-up visit will be performed within 4 weeks (±3 days) from removal of the ICV access device.

### 9.4.5 Method of Assigning Subjects to Treatment Groups

This is a single-arm study. All subjects will receive BMN 190 qow.

#### 9.4.6 Selection of Doses Used in the Study

The planned dose level is 300 mg qow. This dose is based on data from Study 190-201.

The dose level is derived from dose levels used in the TPP1-null dachshund study (Katz, 2014) (Vuillemenot, 2011). Pharmacological effects, including functional improvement and life extension, have been robustly demonstrated in TPP1-null dachshunds at 4 mg and 16 mg dose levels. Human-equivalent doses were calculated by two methods: CSF volume scaling and brain mass scaling. CSF volume for a child aged 2 to 7 years was estimated to be 100 mL, based on normal adult volumes of 125 to 250 mL; the scaling factor is 8-fold for a dachshund CSF volume of 12.5 mL. The human brain on average achieves about 75% of adult mass by age 2 and 100% by age 5 (Giedd, 1996). If adult human brain mass is 1400 g, the range for healthy children aged 2 to 7 years would be 1050 to 1400 g. Given progressive brain atrophy in CLN2 disease patients, an average mass of 1000 g was assumed, yielding a scaling factor of 20-fold based on average dachshund brain mass of 50 g. Since TPP1 activity in brain tissue is more proximally related to CNS lysosomal storage materials, scaling by brain mass is judged to be more predictive of the human therapeutic dose.

The no-observed-adverse-effect level (NOAEL) from nonclinical studies in dachshund was 16 mg, which would correspond to 320 mg in human. Therefore, the starting dose of 30 mg in the preceding study (190-201) is more than 10-fold below the human equivalent of the nonclinical NOAEL.

The clinical experience of BMN 190 for this regimen is justified by the observed safety and tolerability of BMN 190 in Study 190-201 to date.



## 9.4.6.1 Selection of Timing of Dose for Each Subject

A mean CNS half-life of approximately 2 weeks (BMN 190-09-071) suggests biweekly dosing may sustain therapeutic BMN 190 levels in the CNS. BMN 190 concentrations in CSF remained above the lysosomal K<sub>uptake</sub> for approximately 48 hours after single ICV or intrathecal infusions in species with CSF dynamics similar to those in human (Vuillemenot, 2014), (Vuillemenot, 2011), (BMN 190-09-071). In these same species (dog and monkey), CNS distribution of BMN 190 was extensive in many brain regions.

#### 9.4.6.2 Selection of Infusion Volume and Rate

The nonclinical studies in the dachshund and cynomolgus monkey utilized an infusion rate of approximately 5% of the total CSF volume per hour. This was expected to represent a safe infusion rate that would minimize changes in total CSF volume and intracranial pressure. The dachshunds received ICV infusions at a rate of 0.6 mL/hour for 2 hours, while monkeys received 0.88 mL/hour for 3.6 hours. No effects were observed in these studies indicative of safety concerns due to the infusion rate. In the CLN2 patient population, the estimated CSF volume is approximately 100 mL. For the proposed clinical trial, a volume of 10 mL infused over a 4 hour period represents an infusion rate of approximately 2.5% of the total CSF volume per hour, which is approximately half the rate that had no safety effects in the nonclinical studies. Therefore, we expect that 10 mL infused over 4 hours would be safe in CLN2 patients. To date, infusions at parameters listed above in patients in Study 190-201 have shown no safety concerns.

#### 9.4.7 Blinding

This is an open-label study. Study site assessments of safety and clinical severity will be performed without blinding to treatment.

As defined in the Imaging Charter, oversight of MRI evaluation will be performed by independent radiologists at a central imaging facility. The interpreting radiologists and software analysis will be blinded to subject and time on study. All subject-identifying information will be redacted before endpoints are assessed.

Oversight of EEG evaluation will be performed by an independent epileptologist at a central facility. The interpreting epileptologists and software analysis will be blinded to subject and time on study. All subject-identifying information will be redacted before endpoints are assessed.



#### 9.4.8 Prior and Concomitant Medications

Medications (prescription, over-the-counter, and herbal) and nutritional supplements taken during the 30 days before informed consent will be recorded in the eCRF at Screening. At each subsequent visit (or within one week of the Early Termination visit), change in any medication (dosage, frequency, new medication, or cessation) since the previous visit will be recorded in the eCRF

Ongoing medications taken during participation in BMN 190-201 should be recorded in the eCRF. Any concomitant medication added or discontinued during the study should be recorded in the eCRF (or within one week of the Early Termination visit).

It is anticipated that all subjects will be taking anticonvulsants. Subjects may also be taking medications for myoclonus, tremor, agitation, and pain. Investigators will be asked to keep these regimens constant from before the First Dose visit throughout the study, unless changes are required due to lack of efficacy or toxicity.

Use of non-drug therapies such as physical and occupational therapy will also be noted in the eCRF.

### 9.4.9 Treatment Compliance

Study drug will be administered to subjects at the study site by a qualified professional. Date, time, volume, and concentration of each dose must be recorded in the dispensing log as well as on the appropriate eCRF In the event that a dose of study treatment is missed or incomplete, the investigator should record the reason and any other pertinent information on the eCRF as appropriate.

#### 9.5 Investigational Product Accountability

The Investigator or designee is responsible for maintaining accurate records (including dates and quantities) of IP(s) received, subjects to whom IP is dispensed (subject-by-subject dose specific accounting), and IP lost or accidentally or deliberately destroyed. The Investigator or designee must retain all unused or expired study supplies until the study monitor (on-site CRA) has confirmed the accountability data.

# 9.5.1 Return and Disposition of Clinical Supplies

Unused study drug must be kept in a secure location for accountability and reconciliation by the study monitor. The Investigator or designee must provide an explanation for any destroyed or missing study drug or study materials.



Unused study drug may be destroyed on site, per the site's standard operating procedures, but only after BioMarin has granted approval for drug destruction. The monitor must account for all study drug in a formal reconciliation process prior to study drug destruction. All study drug destroyed on site must be documented. Documentation must be provided to BioMarin and retained in the Investigator study files. If a site is unable to destroy study drug appropriately, the site can return unused study drug to BioMarin upon request. The return of study drug or study drug materials must be accounted for on a Study Drug Return Form provided by BioMarin.

All study drug and related materials should be stored, inventoried, reconciled, and destroyed or returned according to applicable state and federal regulations and study procedures.

## 9.6 Dietary or Other Protocol Restrictions

There are no dietary or other protocol restrictions for this study.

#### 9.7 Efficacy and Safety Variables

Although this study is designed to assess safety and tolerability primarily, efficacy will be assessed by impact on disease-specific clinical rating scales. MRI is being assessed as a secondary efficacy variable. Effect on quality of life (QoL), developmental milestones, disease-related biomarkers, EEG, visual acuity, and optical coherence tomography (OCT) will also be explored.

Timing of study assessments is detailed in the Schedule of Events (Table 9.1.1).

# 9.7.1 Primary Efficacy Variables

## 9.7.1.1 Disease-Specific Rating Scales

Disease severity has been evaluated by two CLN2 disease-specific rating scales: the Hamburg Scale (Steinfeld, 2002); (Worgall, 2008) and the Weill Cornell Scale (Dyke, 2012); (Worgall, 2007). Both scales consist of four domains with intrinsic content validity. Within each domain of both scales, a score from 0 to 3 is assigned and overall scores are calculated by summing the four domain scores for a final rating of 0 (severely impaired) to 12 (normal).

Since the domains common to each rating scale, motor (Hamburg) or gait (Weill Cornell) and language, are most relevant to mild to moderate CLN2 disease (Section 9.2), they will be used to assess study eligibility and efficacy (**Appendix 1.**). Timing of post-treatment administration of these rating scales is detailed in Table 9.1.1.

Raters will be identified as qualified practitioners, who have been trained on the definitions and implementation of the CLN2 disease rating scales. All raters at all sites will be required Proprietary and Confidential

17 December 2018



to pass a training session designed to standardize the definitions and scale anchor points across the study, before study ratings take place. Whenever possible, a single rater should evaluate each enrolled patient for the duration of treatment. Further, patient ratings should take place at the same time in the study visit, preferably in the morning before procedures and/or infusion takes place.

Rating scale assessments will be videotaped in a standardized manner across all study sites. The Ratings Assessment Guidelines provide detailed instructions for videotaping. Timing for videotaping of the CLN2 disease scale evaluations is detailed in Table 9.1.1.

### 9.7.2 Secondary Efficacy Variables

### 9.7.2.1 Magnetic Resonance Imaging

All image data will be acquired without contrast on a 1.5 Tesla MRI platform. Study MRIs will include localizer, 3D T1-weighted sagittal, T2-weighted gradient-echo, diffusion-weighted axial and FLAIR axial acquisitions, as specified in the Imaging Charter. Total scanner time is less than 60 minutes and is expected to be accomplished in the majority of subjects with sedation. Volumetric analysis of images will be done by estimating both volume of total cortical grey matter and proportion of the cranial CSF.

Timing of MRIs is detailed in Table 9.1.1.

An MRI scan also should be performed whenever infection or ICV port dysfunction is suspected by the investigator. In this case, according to the Imaging Charter, the MRI should be with or without intravenous contrast with at least T1-weighted axial and sagittal aspects. For suspected meningitis, an MRI of the brain should be performed with and without contrast, according to the Imaging Manual.

# 9.7.3 Exploratory Variables

#### 9.7.3.1 Quality of Life Testing

Quality of life will be assessed using 2 different instruments: the PedsQL™ Measurement Model for Pediatric Quality of Life Inventory (PedsQL) and the CLN2-specific questionnaire.

The age-appropriate assessments for each instrument will be completed for all patients at the timepoints indicated in the Schedule of Events (Table 9.1.1).



# 9.7.3.1.1 PedsQL Measurement Model for Pediatric Quality of Life Inventory

The PedsQL<sup>TM</sup> Generic Core Scales (including both a Parent Report for Toddlers and a Family Impact Module) are designed to measure Quality of Life in children and adolescents. The assessments are brief, practical and developmentally appropriate. The instrument is responsive to clinical change over time (Msall, 2005). The four parent reports cover the ages from 1-12 months, 13-24 months, 2-4 years, and  $\geq$  5 years, and include questions regarding physical, emotional, and social functioning, with school functioning where applicable.

### 9.7.3.1.2 CLN-2 Specific Quality of Life Questionnaire

The CLN2 health related quality of life assessment is a disease specific supplement to the PedsQL using the same format and quantitation. The questionnaire is a novel instrument that was designed in collaboration with patient family and advocacy groups to capture elemental care and quality of life issues in late infantile CLN2 disease.

### 9.7.3.2 Denver II Developmental Screening Test

The Denver II is a revision and update of the Denver Developmental Screening Test. Both tests were designed to monitor the development of infants and preschool-aged children. The tests cover four general functions: personal social (such as smiling), fine motor adaptive (such as grasping and drawing), language (such as combining words), and gross motor (such as walking). Ages covered by the tests range from birth to 6 years.

#### 9.7.3.3 Biomarkers

Blood and CSF will be collected from subjects at the time points indicated inTable 9.1.1 and may be used to evaluate biochemical, molecular, cellular, and genetic aspects relevant to CLN2 disease. CSF and blood will be collected for exploratory biomarker research. Samples will be collected prior to infusion. Exploratory genetic research to study or try to discover genes that are not yet known to be associated with CLN2 disease is optional.

All biomarker samples collected in this study may be used for exploratory biomarker research. In addition, samples collected for other purposes may be used for exploratory use once the primary use has been completed.

#### 9.7.3.4 Electroencephalogram

A standard awake EEG will be recorded within 2 days before each infusion as indicated in Table 9.1.1.

If a clinically significant abnormality is noted, the investigator or designee will evaluate whether study enrollment or continuation is appropriate; a clinically significant abnormality Proprietary and Confidential

17 December 2018



will be recorded under Medical History during Week 1 and as an AE thereafter. Evaluation will be done both locally and by a centralized vendor.

#### 9.7.3.5 Assessments of Visual Acuity

The Preferential Looking Test (PLT) is a method of assessing visual acuity in infants and children with limited cognitive function. The PLT assesses the acuity of children who are unable to identify pictures, shapes, or letters, and is particularly useful in children with physical and/or mental disabilities. The principle of the test is that a young child will choose to look towards an interesting visual stimulus ("target") rather than a plain stimulus. The child is presented with two stimulus fields, one with stripes and the other with a homogeneous gray area of the same average luminance as the striped field. The location of the stripes is randomly alternated. Typically, infants and children will look at the more interesting stripes (if they can detect them) rather than at the blank field. Teller, Keeler, and LEA Grating Acuity Cards have been standardized to assess grating (resolution) visual acuity in infants and nonverbal children using the principles of Preferential Looking.

Other standardized versions of the LEA Test System use symbols or numbers to assess visual acuity in children who do not know how to read the letters of the alphabet that are typically used in an eye chart, but require higher cognitive function than PLT. The symbols are likely to be more useful in the CLN2 patient population. Similarly, the E-Hook or Tumbling E chart has been standardized to use rows of the letter "E" in various orientations. The patient is asked to point to where the limbs of the E are pointing "up, down, left or right." Depending on how far down the chart the patient can "read", his or her visual acuity is quantified.

All subjects will perform PLT. Use of standardized Teller, Keeler, or LEA Grating Cards to perform PLT are all acceptable based on institutional standards and availability of personnel experienced in performing the assessments. The choice of testing materials should be consistent for all patients at each investigational site. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or Tumbling E Vision Test should also be performed during the same assessment using standardized techniques. The choice of additional assessments for higher functioning children (eg, LEA symbol or Tumbling E) should be made based on availability of experienced and qualified personnel to perform the assessment and should remain consistent throughout the study. Whenever possible, all tests of visual acuity should be performed by the same tester.

The tests of visual acuity may be done either before or after drug infusion based on logistical considerations and ease for the subject and study personnel. However, the timing should



remain consistent for all subsequent assessments. Patients must be alert and not influenced by any sedating medications.

# 9.7.3.6 Optical Coherence Tomography

Optical coherence tomography (OCT) is a non-invasive imaging test that uses light waves to take cross-sectional pictures of the retina's layers in order to measure their thickness. These measurements can aid in early detection and treatment for retinal diseases. OCT will be performed locally and should precede infusions. In order to limit the need for sedation to perform this assessment, measurement should be obtained while the subject is also under sedation for MRI acquisition.

OCT images will be collected by BioMarin, to be assessed by BioMarin personnel or designees.

#### 9.7.4 Immunogenicity

Immunogenicity tests will be performed using validated immunogenicity assays on serum and CSF samples. Samples of CSF and serum will be collected for anti-BMN 190 TAb and NAb testing, as detailed in Table 9.1.1. Collection must precede study drug infusion when collected for routine immunogenicity assessments. Baseline blood (serum) samples will be collected at the Study Completion visit in Study 190-201 to obtain a baseline TAb and NAb, every 12 weeks thereafter (Q12W), at the Study Completion or Early Termination visit, at the Device Safety Follow-Up visit, and at the Safety Follow-Up visit. CSF samples will be collected for anti-BMN 190 TAb and NAb testing at the Study Completion visit in Study 190-201 and every 12 weeks thereafter (Q12W). Serum and CSF NAb will be tested at Study Completion Visit in Study 190-201 and at subsequent time points when serum and CSF TAb are positive, respectively. No CSF immunogenicity assessments will be performed at either of the safety follow-up visits.

In the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion). At the Device Safety Follow-Up visit and the Safety Follow-Up visit, serum samples will be collected to assess total IgE, tryptase, and C4.

## 9.7.5 Safety Variables

Safety will be determined from incidence, severity, and relationship to BMN 190 of treatment-emergent AEs/SAEs reported during the study. In addition, weight, height, vital

Proprietary and Confidential

17 December 2018



signs, physical examination, neurologic examination, ECG, standard clinical laboratory blood (chemistry panel and CBC) and urine tests, standard clinical laboratory CSF tests (cell count, protein, glucose, and culture), concomitant medications, and AE/SAEs reported during the study as related to the device will be monitored.

#### 9.7.5.1 Adverse Events

AEs and SAEs will be recorded as defined in Section 10. At each visit, subjects will be asked about new or ongoing AEs since the previous visit.

#### 9.7.5.2 Device Malfunction

For this study, a medical device is defined as the infusion pump and all contact parts (reservoir and catheter, needles, infusion line with filter, extension sets, and syringes) intended to be used for administration of BMN 190. Device malfunctions should be reported following the implantation of the ICV reservoir and catheter. A device malfunction means the failure of a device to meet its performance specifications or otherwise perform as intended. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, should also be returned. For reporting device-related AEs of special interest, please refer to Section 10.3.

## 9.7.5.3 Clinical Laboratory Assessments

Blood and urine samples will be collected for routine clinical laboratory assessments (blood chemistries, hematology, and urinalysis) as detailed in Table 9.1.1.

Any abnormal test result determined clinically significant by the investigator should be repeated until its cause is determined, the value returns to baseline or within normal limits, or the investigator determines the abnormal value was no longer clinically significant.

All abnormal clinical laboratory pages should be initialed and dated by an investigator, along with a comment regarding clinical significance. Each clinically significant laboratory result is to be recorded as medical history at Week 1 and as an AE subsequently.

If known, the diagnosis associated with an abnormality in clinical laboratory results considered clinically significant by the investigator should be recorded on the AE eCRF.



**Table 9.7.5.3.1: Clinical Laboratory Tests** 

| Blood Chemistry | Hematology | Urinalysis |
|----------------------|-------------------------|------------------|
| albumin | hemoglobin | appearance |
| alkaline phosphatase | hematocrit | color |
| ALT (SGPT) | WBC count | pН |
| AST (SGOT) | RBC count | specific gravity |
| direct bilirubin | platelet count | ketones |
| total bilirubin | differential cell count | protein |
| blood urea nitrogen | | glucose |
| calcium | | bilirubin |
| carbon dioxide | | nitrite |
| chloride | | urobilinogen |
| total cholesterol | | hemoglobin |
| C-reactive protein | | |
| creatinine | | |
| creatine kinase | | |
| glucose | | |
| GGT | | |
| LDH | | |
| phosphorus | | |
| potassium | | |
| total protein | | |
| sodium | | |
| uric acid | | |

## 9.7.5.4 Cerebrospinal Fluid Surveillance

Samples of CSF for routine surveillance (cell count with differential, protein, glucose, and culture) will be collected within 30 ( $\pm 5$ ) minutes before every infusion (or within one week of the Early Termination visit), as indicated in Table 9.1.1.

# 9.7.5.5 Other Laboratory Assessments

Subjects who experience an SAE possibly related to BMN 190 or other AE of concern may have additional blood samples drawn to assess immunogenicity, or safety parameters as indicated in Table 9.1.1.



# 9.7.6 Vital Signs, Physical Examinations and Other Observations Related to Safety

### **9.7.6.1** Vital Signs

Vital signs (SBP, DBP, heart rate, respiration rate, and temperature) will be measured as indicated in Table 9.1.1. For every infusion, vital signs (SBP, DBP, heart rate, respiration rate, and temperature) will be measured within 30 (±5) minutes before infusion start (or restart), every 30 (±5) minutes during infusion, 0.5 hours (±5 minutes), 1 hour (±5 minutes), and 4 hours (±15 minutes) after infusion end, and then every 4 hours (±15 minutes) for the next 16 hours. Blood pressure will be measured in the upper arm using an appropriately sized blood pressure cuff. If the patient's blood pressure is abnormal (as compared to site-specific reference ranges), a manual blood pressure will be obtained by a trained healthcare professional.

## 9.7.6.2 Physical Examination

A <u>complete</u> physical examination will be performed as indicated in Table 9.1.1. A complete examination will include general appearance (head, eyes, ears, nose, and throat), cardiovascular, dermatologic, lymphatic, respiratory, gastrointestinal, genitourinary, musculoskeletal, and neurologic systems (level of consciousness, speech, language, cranial nerves, motor strength, motor tone, abnormal movements, reflexes, upper extremity sensation, lower extremity sensations, gait, Romberg, nystagmus, and coordination). Results of the neurologic examination may also be used to assess the efficacy of BMN 190.

A <u>brief</u> physical examination will be performed otherwise, as indicated in Table 9.1.1. A brief examination will include general appearance, cardiovascular, respiratory, neurologic, and gastrointestinal assessments.

Body weight and height assessments should be performed at the timepoints indicated in Table 9.1.1.

Use of an ICV reservoir device for intracerebroventricular drug administration requires that patients be monitored throughout the study for potential infections (high temperature, cough, rash, headache, mental status changes, swelling or drainage in the incision area) and signs of ICV reservoir leakage or failure (swelling of skin around reservoir site, difficulty with CSF extraction, erythema of the scalp, bulging of reservoir device, or extravasation of fluid on infusion).

The investigator will evaluate the patency, location, and skin integrity of the reservoir at each study drug administration. The investigator will check for scalp edema, erythema or skin breakdown at the site of the reservoir prior to infusion. Patency will be assessed during



pre-infusion sampling and again at the time of infusion. Difficulty in obtaining the required volume of CSF necessary for pre-infusion samples or signs of ICV reservoir leakage (swelling of skin around reservoir site, erythema of the scalp, bulging of reservoir device, or extravasation of fluid) will prompt further evaluation of the reservoir for failure prior to continuing with infusion. Additional surgical consultation including surgery may be required to revise or replace the device. Material degradation of the ICV device reservoir has occurred after approximately 105 perforations of the ICV device in benchtop testing, and has been observed in clinical trials with approximately 4 years of BMN 190 administration. Access device replacement should be considered prior to 4 years of regular administration of BMN 190; with the decision made on an individual subject level based on the medical judgment of the Investigator. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, should also be returned.

Clinically significant abnormalities noted during physical examination will be recorded under Medical History at Week 1 or as AEs thereafter.

# 9.7.6.3 Electrocardiogram

For at least one infusion of BMN 190 (and preferably the next infusion), continuous ECG monitoring (3- or 5-lead) will be performed for all subjects. The ECG should begin 15 (±5 minutes) prior to infusion start, continue through infusion of BMN 190, and end after infusion of flushing solution. If a 12-lead ECG is required during this time, continuous monitoring should be interrupted in order to obtain the 12-lead ECG.

A standard ECG (12-lead), including heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities, will be performed 30 (±5) minutes after infusion end at the first infusion and every 24 weeks thereafter. In patients with present or past bradycardia, conduction disorders, or with structural heart disease, an ECG will be performed within 30 minutes before the start of infusion (±5 minutes), at 2 hours (±15 minutes) during infusion, 30 (±5) minutes after infusion end, and 12 hours (±3 hours) after infusion end for each study drug infusion.

If a clinically significant abnormality is noted, the investigator or designee will evaluate whether study enrollment or continuation is appropriate; a clinically significant abnormality will be recorded under Medical History during Week 1 and as an AE thereafter.



# 9.7.6.4 Pregnancy Testing

A pregnancy test will be performed during the Screening period on female subjects of childbearing potential.

A female subject judged by the investigator to be of childbearing potential will be tested for pregnancy with a urine pregnancy test; additional urine tests will be performed during the study whenever pregnancy is in question. A serum pregnancy test will be performed if a urine test result is positive or equivocal.



## 10 REPORTING ADVERSE EVENTS

#### 10.1 Adverse Events

For this protocol, a reportable adverse event (AE) is any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a patient administered the study-drug or other protocol-imposed intervention, regardless of attribution. This includes the following:

- AEs not previously observed in the subject that emerge during the course of the study.
- Pre-existing medical conditions judged by the Investigator to have worsened in severity or frequency or changed in character during the study.
- Complications that occur as a result of non-drug protocol-imposed interventions (e.g., AEs related to screening procedures, medication washout, etc.).

An adverse drug reaction is any AE for which there is a reasonable possibility that the study-drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study-drug and the AE.

Whenever possible, it is preferable to record a diagnosis as the AE term rather than a series of terms relating to a diagnosis.

All AEs/ SAEs/ adverse events of special interest (AEOSIs) / pregnancies will be recorded starting after the first dose of study drug in Study 190-202. Reporting of AEs/SAEs / AEOSIs/ pregnancies will continue until 6 months after either the last administration of study drug or the Early Termination visit. The 6-month Safety Follow-Up Visit will be waived for subjects who begin receiving study drug in another BioMarin-sponsored study or registry within this 6-month period. For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug. For subjects who enroll into another BioMarin-sponsored study or registry, AE/SAE / AEOSI/ pregnancy reporting is as follows:

- The 190-202 reporting period for new onset AEs/SAEs, pregnancies, and device-related events ends when the subject receives the first dose of study drug under the new study or registry.
- Ongoing AEs related to study drug will be followed until resolution under this study.
- All ongoing SAEs, pregnancies, and device-related events will be followed until resolution under this study.



• Events that started in this study and worsen after first the dose of study drug in the new study or registry will be captured as a new event under the new study.

Criteria for determining and reporting SAEs is provided in Section 10.2.

For this study, a medical device is defined as the infusion pump and all contact parts components required for infusion (reservoir and catheter, needles, infusion line with filter, extension sets, and syringes) intended to be used for administration of BMN 190. Adverse events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be entered into the device AE/SAE eCRF and the device report form and reported to BioMarin Pharmacovigilance (BPV) within 24 hours by entering the event information via EDC and completing the study specific device report form(s). Prophylactic replacement of the ICV must be reported as a device related event. The reporting period for device-related events is the same as the reporting period for all AEs and SAEs; if the device is removed prior to the 6 month safety follow-up visit, the follow-up safety reporting period for device-related events is 4 weeks from the removal of the device.

The Investigator should follow all unresolved AEs until the events are resolved or stabilized, the patient is lost to follow-up, or it has been determined that the study treatment or participation is not the cause of the AE. Outcome of AEs (with dates) should be documented on the appropriate eCRF page(s) and in the patient's medical record.

The Investigator responsible for the care of the patient or medically qualified designee will assess AEs for severity, relationship to study-drug, and seriousness (see Section 10.2 for SAE definition). Severity (as in mild, moderate or severe headache) is not equivalent to seriousness, which is based on patient/event outcome or action criteria usually associated with events that pose a threat to a patient's life or functioning.

#### 10.1.1.1 Seriousness

The investigator will assess if an AE should be classified as "serious" based on the seriousness criteria enumerated in Section 10.2. Seriousness serves as a guide for defining regulatory reporting obligations.

#### **10.1.1.2** Severity

The severity of each AE will be assessed using the defined categories in Table 10.1.1.2.1.

The Investigator will determine the severity of each AE and SAE and AEoSI using the NCI CTCAE v4. Adverse events that do not have a corresponding CTCAE term will be assessed according to the general guidelines for grading used in the CTCAE v4 as stated below.



Table 10.1.1.2.1: Adverse Event Grading (Severity) Scale

| Grade | Description | |
|---|---|---|
| 1 | Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | |
| 2 | Moderate: minimal, local or noninvasive intervention indicated; limiting age-<br>appropriate instrumental activities of daily living (ADL) <sup>a</sup> | |
| 3 | Severe or medically significant but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL <sup>b</sup> | |
| 4 | Life threatening: urgent intervention indicated | Grade 4 and 5 AEs |
| 5 | Death related to AE | should always be reported as SAEs |

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to the following examples: preparing meals, shopping for groceries or clothes, using the telephone, managing money.

# **10.1.1.3** Causality

The Investigator will determine the relationship of an AE to the study drug and will record it on the source documents and AE CRF. To ensure consistency of causality assessments, Investigators should apply the guidance in Table 10.1.1.3.1.

<sup>&</sup>lt;sup>b</sup> Self-care ADL refer to the following examples: bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, not bedridden.



**Table 10.1.1.3.1: Causality Attribution Guidance** 

| Relationship | Description |
|---|---|
| Not Related | Exposure to the IP has not occurred |
| | OR |
| | <ul> <li>The administration of the IP and the occurrence of the AE are not<br/>reasonably related in time</li> </ul> |
| | OR |
| | • The AE is considered likely to be related to an etiology other than the use of the IP; that is, there are no facts, evidence, or arguments to suggest a causal relationship to the IP. |
| Related | • The administration of the IP and the occurrence of the AE are reasonably related in time |
| | AND |
| | <ul> <li>The AE could possibly be explained by factors or causes other than<br/>exposure to the IP</li> </ul> |
| | <u>OR</u> |
| | <ul> <li>The administration of IP and the occurrence of the AE are reasonably<br/>related in time</li> </ul> |
| | AND |
| | <ul> <li>The AE is more likely explained by exposure to the IP than by other<br/>factors or causes.</li> </ul> |

Factors suggestive of a causal relationship could include (but are not limited to):

- Plausible temporal relationship
- Absence of alternative explanations
- Rarity of event in a given patient or disease state
- Absence of event prior to study drug exposure
- Consistency with study product pharmacology
- Known relationship to underlying mechanism of study drug action
- Similarity to adverse reactions seen with related drug products
- Abatement of AE with discontinuation of study drug, and/or recurrence of AE with reintroduction of study drug

The investigator's assessment of causality for individual AE reports is part of the study documentation process. Regardless of the Investigator's assessment of causality for individual AE reports, the Sponsor will promptly evaluate all reported SAEs against cumulative product experience to identify and expeditiously communicate (in compliance



with applicable regulations) possible new safety findings to investigators and applicable regulatory authorities.

#### 10.2 Serious Adverse Events

A serious adverse event (SAE) is any untoward medical occurrence that at any dose meets one or more of the following criteria:

- Is fatal
- Is life threatening

Note: Life-threatening refers to an event that places the patient at immediate risk of death. This definition does not include a reaction that, had it occurred in a more severe form, might have caused death.

- Requires or prolongs inpatient hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly or birth defect in the child or fetus of a patient exposed to IP prior to conception or during pregnancy
- Is an important medical event or reaction that based on medical judgment, may jeopardize the patient or require intervention to prevent one of the above consequences (e.g., anaphylaxis).

All adverse events that do not meet any of the criteria for SAEs should be regarded as non-serious AEs.

The reporting period for SAEs begins after the first dose of study drug in Study 190-202 and continues until 6 months after either the last administration of study drug or the Early Termination visit. The 6-month Safety Follow-Up Visit will be waived for subjects who begin receiving study drug in another BioMarin-sponsored study or registry within this 6-month period. Refer to Section 10.1 for additional information regarding SAE reporting for these subjects. For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug. If a subject is discontinued from the study prematurely, SAEs will be recorded at the Early Termination visit.

Exclusions to SAE reporting include planned hospitalization for a study procedure or elective surgery before study enrollment. Events that occur as a result of these hospitalizations or surgeries that meet SAE reporting requirements are reportable to BPV within 24 hours.



All SAEs, including device-related events, whether or not considered related to study drug, must be reported within 24 hours of the site becoming aware of the event. SAEs will be reported via eCRF to BPV. If the eCRF system is not available the SAE must be reported on the study specific SAE report form and entered into eCRF when possible. Device and device component related events will also require completion of the study specific Device Report form and must be submitted to BPV within 24 hours. Investigators should not wait to collect information that fully documents the event before notifying BPV of an SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that investigators submit any information requested by BioMarin as soon as it becomes available. The Sponsor is responsible for identifying, preparing, and reporting all suspected unexpected serious adverse reactions (SUSARs) to the relevant competent authorities, ethics committees, and investigators in accordance with requirements identified in the Clinical Trials Regulations.

The investigator should follow any unresolved SAE until the event is resolved or stabilized, the subject is lost to follow-up, or it has been determined that study treatment or participation is not the cause of the SAE. Resolution of SAEs (with dates) should be documented in the eCRF and in the subject's medical record.

For some SAEs, BioMarin may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details (e.g., hospital discharge summary, consultant report, or autopsy report) deemed necessary to appropriately evaluate the SAE report.

At the last scheduled visit, the investigator should instruct each subject to report, to the investigator and/or to BPV directly, any subsequent SAE that the subject's personal physician believes might be related to prior study treatment.

The investigator should notify BioMarin of any death or SAE occurring any time after a subject has discontinued or terminated study participation if the investigator believes the death or SAE may have been related to prior study treatment. BioMarin should also be notified if the investigator becomes aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject who participated in this study.

Reporting of SAEs to the IRB or IEC will be done in compliance with the standard operating procedures and policies of the IRB or IEC and with applicable regulatory requirements. Adequate documentation must be obtained by BioMarin showing that the IRB or IEC was properly and promptly notified as required.



## 10.3 Adverse Events of Special Interest

AEOSIs may be assessed by the Investigator as serious or non-serious. AEOSIs for this study include status epilepticus, hydrocephalus (communicating and noncommunicating), meningitis, unexpected rapid decline on CLN2 disease scale not attributable to other causes, hypersensitivity, all device-related events (e.g., infection, malfunction with an associated AE such as leaking reservoir or a problem that ends the administration of study drug for that visit, etc.), cardiovascular events, ECG adverse events, and any temporally-related adverse event, defined as events which occur within 24 hours of BMN 190 infusion; any of these events must be reported to BPV using the appropriate eCRF, irrespective of severity, seriousness, or causality within 24 hours of a study site awareness. Device-related events (eg, infection, malfunction with an associated AE, such as leaking reservoir or a problem that ends the administration of study drug for that visit) require the completion of the Device Event Report Form in addition to eCRF reporting. All removed or replaced implantable ICV devices must be reported as device-related events and should be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual), except for infusion pumps, should also be returned.

Subjects will be monitored during and following infusion (Section 9.4.4). Any AE, including anaphylaxis and other hypersensitivity or allergic reaction, occurring within 24 hours after the start or restart of a BMN 190 infusion, regardless of investigator assessment of study drug relationship, will be assessed as a hypersensitivity reaction. As stated above, the investigator must report the event to BPV using the appropriate eCRF within 24 hours of a hypersensitivity reaction. The investigator is encouraged to discuss with the BioMarin medical monitor all AEOSIs as defined above.

#### 10.4 Procedures for Recording Adverse Events

# 10.4.1 Recording Adverse Events on a eCRF

Investigators should use precise medical terminology when recording AEs or SAEs. Avoid colloquialisms and abbreviations.

Record only one diagnosis, sign, or symptom per event field on the AE eCRF (e.g., nausea and vomiting should not be recorded in the same entry, but as 2 separate entries).

In order to classify AEs and diseases, preferred terms will be assigned by the Sponsor to the original terms entered on the eCRF, using MedDRA (Medical Dictionary for Regulatory Activities) terminology.



# 10.4.2 Diagnosis versus Signs and Symptoms

Using accepted medical terminology, enter the diagnosis (if known). If not known, enter sign(s) and/or symptom(s). If a diagnosis subsequently becomes available, then this diagnosis should be entered on the AE eCRF, replacing the original entries where appropriate.

## 10.4.3 Adverse Events Occurring Secondary to Other Events

In general, AEs occurring secondary to other events (e.g., cascade events) should be identified by their primary cause. For example, if severe diarrhea is known to have resulted in dehydration, it is sufficient to record only diarrhea as an AE or SAE on the eCRF. However, medically important events that may be linked and/or separated in time should be recorded as independent events on the eCRF. For example, if severe hemorrhage leads to renal failure, both events should be recorded separately on the eCRF.

#### 10.4.4 Persistent or Recurrent Adverse Events

A persistent AE is one that extends continuously, without resolution, between patient evaluation time points with no change in severity. For non-serious AEs, if the severity changes (increases or decreases), a new AE should be entered on the AE eCRF (in which case it should be recorded again on the AE eCRF). AEs characterized as intermittent require documentation of onset and duration of each episode.

A recurrent AE is one that occurs and resolves between patient evaluation time points, but then subsequently recurs (such as seizures). Each recurrence of the AE should be recorded on the AE eCRF.

#### 10.4.5 Abnormal Laboratory Values

Laboratory test results will be recorded on the laboratory results pages of the eCRF, or appear on electronically produced laboratory reports submitted directly from the central laboratory, if applicable.

Any laboratory result abnormality fulfilling the criteria for a SAE should be reported as such, in addition to being recorded as an AE in the eCRF.

A clinical laboratory abnormality should be documented as AE if **any** of the following conditions is met:

Accompanied by clinical symptoms



- Leading to a change in study medication (e.g., dose modification, interruption or permanent discontinuation)
- Requiring a change in concomitant therapy (e.g., addition of, interruption of, discontinuation of, or any other change in a concomitant medication, therapy or treatment).
- The laboratory abnormality is not otherwise refuted by a repeat test to confirm the abnormality
- The abnormality suggests a disease and/or organ toxicity
- The abnormality is of a degree that requires active management (e.g., change of dose, discontinuation of study drug, more frequent follow-up assessments, further diagnostic investigation, etc.)

This applies to any protocol and non-protocol specified safety and efficacy laboratory result from tests performed after the first dose of study medication that falls outside the laboratory reference range and meets the clinical significance criteria.

This does not apply to any abnormal laboratory result that falls outside the laboratory reference range but that does not meet the clinical significance criteria (these will be analyzed and reported as laboratory abnormalities), those that are considered AEs of the type explicitly exempted by the protocol, or those which are a result of an AE that has already been reported.

### **10.4.6 Pre-existing Conditions**

A pre-existing condition is one that is present at the start of the study. Such conditions should be recorded as medical history on the appropriate eCRF. Ongoing AEs from Study 190-201 will be recorded as medical history in Study 190-202 on the appropriate eCRF.

A pre-existing condition should be recorded as an AE or SAE during the study **only** if the frequency, intensity, or character of the condition worsens during the study period. It is important to convey the concept that a pre-existing condition has changed by including applicable language in the verbatim description of the event (e.g., *more frequent* headaches).

# 10.4.7 General Physical Examination Findings

At screening, any clinically significant abnormality should be recorded as a pre-existing condition (refer to Section 9.7.6.2). During the study, any new clinically significant findings and/or abnormalities discovered on physical examination that meet the definition of an AE (or an SAE) must be recorded and document as an AE or SAE on the AE eCRF.



## 10.4.8 Hospitalization, Prolonged Hospitalization, or Surgery

Any AE that results in hospitalization or prolonged hospitalization should be documented and reported as an SAE unless specifically instructed otherwise in this protocol (refer to Section 10.2).

There are some hospitalization scenarios that do not require reporting as an SAE when there is no occurrence of an AE. These scenarios include planned hospitalizations or prolonged hospitalizations to:

- Perform a protocol-mandated procedure (excludes prophylactic ICV replacement)
- Undergo a diagnostic or elective surgical procedure for a pre-existing medical condition that has not changed
- Receive scheduled therapy (study drug or otherwise) for the study indication

#### **10.4.9 Deaths**

All deaths that occur during the AE reporting period (refer to Section 10.1), regardless of attribution, will be recorded on the AE eCRF and expeditiously reported to the Sponsor (in compliance with applicable regulations) as an SAE. If the death is assessed as related the device (or any of its components), the study specific Device Report Form must be completed and submitted to BPV within 24 hours of the site becoming aware of the event.

When recording a death, the event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the eCRF. If the cause of death is unknown and cannot be ascertained at the time of reporting, record "Unexplained Death" on the eCRF. If the death is attributed to progression of the disease or condition being studies, record "Disease Progression" as the SAE term on the eCRF.

#### 10.4.10 Pregnancy

Although not an AE per se, pregnancy in either a patient or the partner of a patient taking trial medication should be expeditiously reported to BPV in compliance with applicable regulations to facilitate outcome monitoring by the Sponsor. Refer to Section 10.1 for pregnancies reporting period.

Pregnancy in a patient or partner should be reported within 24 hours of the site becoming aware of the pregnancy by completing the Pregnancy eCRF and submitting to BPV. In addition, pregnancy in a patient is also reported on the End of Study eCRF. The Investigator must make every effort to follow the patient through resolution of the pregnancy (delivery or termination) and to report the resolution on the Pregnancy Follow-up



Form eCRF. In the event of pregnancy in the partner of a study patient, the Investigator should make every reasonable attempt to obtain the woman's consent for release of protected health information.

Abortion, whether therapeutic or spontaneous, should always be classified as an SAE (as the Sponsor considers these to be medically significant), recorded on the AE eCRF, and expeditiously reported to the Sponsor as an SAE in compliance with applicable regulations.

## **10.4.11** Reporting Requirements

#### 10.4.11.1 Expedited Reporting Requirements

All SAEs AEOSIs, and pregnancies that occur during the course of the AE Reporting Period, whether or not considered related to study drug, must be reported via eCRF to BPV within 24 hours of the site becoming aware of the event. If the eCRF system is not available the SAE must be reported on the study specific SAE report form and entered into eCRF when possible. If the AE is assessed as related to the device (or any of its components), the study specific Device Report form must be completed and submitted via email/FAX within 24 hours of the site becoming aware of the event. Investigators should not wait to collect information that fully documents the event before notifying BPV of an SAE. BioMarin may be required to report certain SAEs to regulatory authorities within 7 calendar days of being notified about the event; therefore, it is important that Investigators submit any information requested by BioMarin as soon as it becomes available. The reporting period for SAEs begins after informed consent is obtained and continues until 6 months following either the last administration of study drug or study discontinuation/termination, whichever is longer (also see Section 10.2).

## **10.5** Urgent Safety Measures

The regulations governing clinical trials state that the sponsor and Investigator are required to take appropriate urgent safety measures to protect subjects against any immediate hazards that may affect the safety of subjects, and that the appropriate regulatory bodies should be notified according to their respective regulations. According to the European Union (EU) Clinical Trial Directive 2001/20/EC, "...in the light of the circumstances, notably the occurrence of any new event relating to the conduct of the trial or the development of the investigational medicinal product where that new event is likely to affect the safety of the subjects, the sponsor and the Investigator shall take appropriate urgent safety measures to protect the subjects against any immediate hazard. The sponsor shall forthwith inform the competent authorities of those new events and the measures taken and shall ensure that the



IRB/EC/REB is notified at the same time." The reporting period for these events which may require the implementation of urgent safety measures is the period from the time of signing of the ICF through the completion of the last study visit or at the ETV.

Investigators are required to report any events which may require the implementation of urgent safety measures to BioMarin within 24 hours.

Examples of situations that may require urgent safety measures include discovery of the following:

- Immediate need to revise the IP administration (i.e., modified dose amount or frequency not defined in protocol).
- Lack of study scientific value, or detrimental study conduct or management.
- Discovery that the quality or safety of the IP does not meet established safety requirements.

## 10.6 BioMarin Pharmacovigilance Contact Information

Contact information for BioMarin Pharmacovigilance is as follows:

BioMarin Pharmaceutical Inc.

Address 105 Digital Drive

Novato, CA 94949

Phone: (415) 506-6179 Fax: (415) 532-3144

E-mail: drugsafety@bmrn.com

The investigator is encouraged to discuss with the BioMarin medical monitor any AE for which the issue of seriousness is unclear or questioned. The investigator is also encouraged to discuss with the BioMarin medical monitor all events of special interest referenced in Section 10.3. Contact information is as follows:

Name: PI
Address: 105 Digital Drive

Novato, CA 94949 USA

Phone: PI E-mail: PI



#### 11 APPROPRIATENESS OF MEASUREMENTS

#### 11.1 Natural History Studies

Two ongoing prospective natural history studies of CLN2 disease (Weill Cornell Medical Center and University Medical Center, Hamburg, Germany) continue to provide evidence that rating scale scores change in a predictable manner with increasing disease duration (Steinfeld, 2002); (Worgall, 2007).

The Weill Cornell database comprises approximately 45 patients with genetically diagnosed CLN2 disease and includes Weill Cornell Scale scores, some modified Hamburg Scale scores, and MRI data, which has been shared with BioMarin (Crystal, 2004). Approximately half the patients have two assessments 2 weeks to 16 months apart.

The Hamburg registry includes both retrospective and prospective data from approximately 30patients with CLN2 disease with scoring of 6-month periods from birth to 8-10 years of age. All participants are genetically diagnosed; data include Hamburg Scale scores, neurologic and cardiologic examinations, ophthalmology testing, routine clinical pathology, volumetric MRI, EEG, ECG, and echocardiogram. Although clinical data have accrued for up to 10 years, MRI data collection started in 2009 and these data have been shared with BioMarin (A Schulz and A Kohlschütter, Hamburg).

BioMarin plans to construct a combined database with demographics, genotype, CLN2 disease rating scale scores, and supporting clinical data from both natural history studies. MRI imaging data may be included, if feasible. Patients will have scores for the Weill Cornell Scale, the Hamburg Scale, or both scales. BioMarin will investigate the feasibility of imputing both CLN2 disease scores for all patients using clinical data to derive the missing domains. At minimum, there are two shared domains in the two CLN2 disease scales (gait/motor and language), which might be combined.

The natural history data will be used to (1) better understand the performance properties of the two CLN2 disease scales, (2) evaluate correlations between the scales and independent clinical measures, (3) identify other potential clinical outcomes that are relevant and change with disease duration and severity, and (4) generate the group of untreated patients that will be used for comparison to the treated study population of Study 190-201 and Study 190-202.

## 11.2 Disease-Specific Rating Scales

Disease severity has been evaluated by two CLN2 disease-specific rating scales: the Hamburg Scale (Steinfeld, 2002); (Worgall, 2008) and the Weill Cornell Scale (Dyke, 2012);



(Worgall, 2007). Both consist of 4 domains (Appendix 1), each of which has intrinsic high content validity. Within each domain, a score from 0 to 3 is assigned and overall scores are calculated by summing the four domain scores for a final rating of 0 (severely impaired) to 12 (normal).

A modified form of that scale, the Modified Hamburg Scale, demonstrated statistically significant slowing of neurologic decline in subjects receiving gene therapy intervention when compared with decline among control subjects (Worgall, 2008). A second CLN2 disease rating scale, the Weill Cornell Scale (Dyke, 2012); (Worgall, 2007), has also been used to evaluate CLN2 disease severity with highly comparable results.

Although all 4 domains of each rating scale will be completed (Appendix 1), the 2 domains common to both, motor (Hamburg) or gait (Weill Cornell) and language, are expected to be most useful for this study. The remaining 2 domains in each rating scale (Appendix 1) are less likely to be informative for this study. In the Hamburg Scale, vision and seizure domains are weak indicators of disease severity since (1) ICV-delivered BMN 190 is not expected to penetrate the posterior ocular chamber to reach the optic nerve, and (2) seizures managed with pharmacotherapy preclude measurable change in response to treatment, respectively. Similarly, in the Weill Cornell Scale, feeding and myoclonus domains are not ideal for this study since (1) the feeding score may be misleading since a feeding tube often is inserted merely to facilitate care and, thus, does not reflect disease severity necessarily, and (2) the myoclonus score may be misleading since presence or absence of different movement disorders (chorea, tremor, athetosis) are presumed to reflect disease severity.

Because of practical (limited number of available patients) and ethical (neurosurgery in children with fatal neurologic disease) concerns, this study design cannot involve contemporaneous, matched, randomized, blinded, or untreated control subjects (Arkin, 2005); (Crystal, 2004). Therefore, changes in CLN2 disease scale scores will be compared with historical data from at least two registries (Weill Cornell Medical Center in New York and University Medical Center in Hamburg, Germany).

# 11.3 Magnetic Resonance Imaging

As patients progress from mild to severe CLN2 disease, MRI has indicated progressive loss of cortical volume and ventricular enlargement (Worgall, 2007). By late CLN2 disease stages, despite their young age, these patients exhibit substantial atrophy predominantly in the cortical grey matter, comparable to that in elderly people with severe Alzheimer's disease. Magnetic resonance spectroscopy (MRS) in patients with CLN2 disease has demonstrated reduced neuronal N-acetyl-aspartate (NAA), reduced NAA/creatine metabolite



ratios, and increased myoinositol/creatine rations when compared with healthy individuals (Seitz, 1998).

Of all 10 MRI measurements examined to quantitate CLN2 disease progression (Worgall, 2007), ventricular volume or percentage ventricular volume correlated most strongly with age (r²=0.67-0.87), duration of disease (r²=0.71-0.79), and severity on clinical rating scales (r²=0.56-0.76), suggesting that the measurement of ventricular volumes may be the most relevant and sensitive MRI measurement of disease progression. Based on these data, MRI measures of atrophy are more strongly correlated with disease progression than are MRS measures of neuronal viability.

In nonclinical CLN2 disease studies with TPP1-null dachshunds, MRI measurement of ventricular volume enlargement was reduced with BMN 190 treatment (Katz, 2014). Therefore, this first clinical study of CLN2 disease will include MRI measurement of ventricular volume.



#### 12 STUDY PROCEDURES

#### 12.1 Screening/Baseline

Baseline values will be recorded at first infusion, Week 1 Day 1 of Study BMN 190-202. These values will serve as the Baseline values for Study 190-202.

A 2-week Screening period will occur beginning with the Week 47 visit of Study 190-201. During this period, after the nature of the study has been explained, written informed consent by parent or authorized legal guardian must be obtained prior to any research-related procedures.

The following procedures will be performed during the Screening Period:

- Informed consent/assent
- Criteria for study entry
- Pregnancy testing

## 12.2 Treatment Visit(s)

#### 12.2.1 Every Visit (every 2 weeks $\pm$ 3 days)

Treatment visits should occur every 2 weeks ( $\pm$  3 days) during the study. Every effort should be made to ensure that treatment visits occur on a fixed schedule every 2 weeks starting from the first treatment visit in the study.

The first treatment visit will occur at Week 1 of Study 190-202. During every visit, the following procedures will be performed:

- Medical history (Week 1 only)
- Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate)
- For at least one infusion of BMN 190 (and preferably the next infusion), continuous ECG monitoring (3- or 5-lead) will be performed for all subjects. The ECG should begin 15 (± 5 minutes) prior to infusion start, continue through infusion of BMN 190, and end after infusion of flushing solution. If a 12-lead ECG is required during this time, continuous monitoring should be interrupted in order to obtain the 12-lead ECG.
- ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities) 30 (±5) minutes after infusion end for the first infusion. In patients with present or past bradycardia, conduction disorders, or with structural heart disease, an ECG will be performed within 30 minutes before the start of infusion (±5 minutes), at 2 hours (±15 minutes) during infusion, 30 (±5) minutes after infusion end, and 12 hours (±3 hours) after infusion end.



- CSF surveillance (cell count, protein, glucose, and culture) (not required for Week 1, as will be done at the Study Completion visit in Study 190-201)
- Assessment of device patency and device site infection
- Brief physical examination (not required for Week 1, as a complete physical examination will be done at the Study Completion visit in Study 190-201)
- AE assessment (investigator may collect additional blood samples for safety or immunogenicity testing for any AE of concern) (not required for Week 1, as will be done at the Study Completion visit in Study 190-201)
- Concomitant medication assessment (not required for Week 1, as will be done at the Study Completion visit in Study 190-201)
- Study drug infusion
- Telephone call to parent/guardian approximately 48 hours after having been discharged from the visit

#### **12.2.2** Every 8 Weeks

Every 8 weeks (± 3 days) (Weeks 9, 17, 25, 33, 41, 49, 57, 65, 73, 81, 89, 97, 105, 113, 121, 129, 137, 145, 153, 161, 169, 177, 185, 193, 201, 209, 217, 225, 233), the following procedures will be performed:

• CLN2 disease rating scales

#### **12.2.3** Every **12** Weeks

Every 12 weeks (± 3 days) (Weeks 13, 25, 37, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, 169, 181, 193, 205, 217, 229), the following procedures will be performed:

- CSF/serum for immunogenicity
- Visual acuity testing
  - O All subjects will undergo Preferential Looking Testing every 12 weeks. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or E Hook (or Tumbling E) Vision Test should also be performed during the same assessment. Visual acuity testing can be performed either before or after the infusion (± 3 days), but should be performed at a time (relative to infusion) that can be repeated consistently between study visits. The subject must not be sedated at the time of visual acuity testing.
- Blood/urine for clinical lab tests
- Neurological examination
|----------|---------------------|---------|

### 12.2.4 Every 24 Weeks

Every 24 weeks (± 3 days) (Weeks 25, 49, 73, 97, 121, 145, 169, 193, 217), the following procedures will be performed:

- Height and body weight assessment
- CLN2 disease rating scales with videotaping
- ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities) 30 (±5) minutes after infusion end
- EEG, standard awake
- MRI (±4-week window is allowed for this assessment and may be performed at the same time as a scheduled infusion)
- CSF/blood for disease-related biomarkers
- Optical coherence tomography
- CLN2-specific QoL questionnaire
- PedsQL
- Denver II Developmental Scale

### 12.2.5 Every 48 Weeks

The following procedures should be performed every 48 weeks during the study:

• Complete physical examination

### 12.3 Study Completion or Early Termination Visit

The Study Completion visit will occur 2 weeks (± 3 days) after the last dose of BMN 190 (Week 239), or within 1 week of early study termination. At the Study Completion or Early Termination visit, the following procedures will be completed:

- Hamburg and Weill Cornell CLN2 disease rating scales (Appendix 1) videotaped
- ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities)
- EEG (standard awake)
- MRI (±4-week window is allowed for this assessment and may be performed at the same time as a scheduled infusion)
- CSF surveillance (cell count, protein, glucose, and culture)
- CSF and blood for biomarker assays

|----------|---------------------|---------|

- CSF and serum for immunogenicity (TAb; NAb if TAb positive)
- Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate)
- Complete physical examination
- Height and body weight assessment
- Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis)
- PedsQL
- Visual acuity testing
  - All subjects will undergo Preferential Looking Testing. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or E Hook (or Tumbling E) Vision Test should also be performed during the same assessment.
- Optical coherence tomography
- CLN2-specific QoL questionnaire
- Denver II Developmental scale
- Neurological examination
- AE assessment (investigator may collect additional blood samples for safety or immunogenicity testing for any AE of concern)
- Concomitant medication assessment

Following the Study Completion Visit or Early Termination Visit, subjects who will not be continuing to receive BMN 190 in another setting (e.g., commercial use, participation in a registry, participation in another BMN 190 clinical study, etc.) should have their ICV access device removed. Removal of the device should occur no more than 4 weeks after the Study Completion Visit or ETV. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, should also be returned.

### 12.4 Device Safety Follow-Up

Subjects will return to the study site 4 weeks (±3 days) after removal of the ICV access device, when the following procedures will be completed:

- CLN2 disease rating scales (videotaping not required)
- Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate)

|----------|---------------------|---------|

- Brief physical examination (including close examination of the former device site to check for signs of infection, etc.)
- Neurological examination
- Serum for immunogenicity (TAb)
- Serum for total IgE, C4, and tryptase
- Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis)
- AE assessment (investigator may collect additional blood samples or CSF by lumbar puncture for safety or immunogenicity testing for any AE of concern), including ongoing events at the time of the last dose or new events related to study drug.
- Concomitant medication assessment

The 4-week Device Safety Follow-Up Visit will be waived for subjects who do not undergo device removal because they will be continuing to receive BMN 190 in another setting (e.g., commercial use, participation in a registry, participation in another BMN 190 clinical study, etc.).

# 12.5 Safety Follow-Up

Subjects will return to the study site 6 months after the last study treatment, when the following procedures will be completed:

- CLN2 disease rating scales (videotaping not required)
- ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities)
- EEG (standard awake)
- Serum for immunogenicity (TAb)
- Serum for total IgE, C4, and tryptase
- Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate)
- Complete physical examination
- Height and body weight assessment
- Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis)
- AE assessment (investigator may collect additional blood samples for safety or immunogenicity testing for any AE of concern), including ongoing events at the time of the last dose or new events related to study drug.
- Concomitant medication assessment

|----------|---------------------|---------|

The 6-month Safety Follow-Up Visit will be waived for subjects who receive study drug in another BioMarin-sponsored study or registry within this 6-month period.

## 12.6 Study Termination

The study will end after the last subject completes the last Safety Follow-Up visit. BioMarin reserves the right to discontinue the study any time for clinical or administrative reasons and to discontinue participation of an individual investigator or site for clinical or administrative reasons, including, but not limited to, poor enrollment or noncompliance with procedures of the protocol or GCP. In addition, the study may be terminated if, in the opinion of BioMarin, the safety of the study subjects may be compromised.



# 13 DATA QUALITY ASSURANCE

BioMarin personnel or designees will visit the study site prior to initiation of the study to review with the site personnel information about the IP, protocol and other regulatory document requirements, any applicable randomization procedures, source document requirements, eCRFs monitoring requirements, and procedures for reporting AEs, including SAEs.

At visits during and after the study, a CRA will monitor the site for compliance with regulatory documentation, with a focus on accurate and complete recording of data on eCRFs from source documents, adherence to protocol, randomization (if applicable), SAE reporting and drug accountability records.

The designated clinical data management group will enter or transfer eCRF data into a study database.

Data quality control and analysis will be performed by BioMarin or a designee, based on a predefined analysis plan.



#### 14 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

Because the completeness of the data affects the integrity and accuracy of the final study analysis, every effort should be made to ensure complete, accurate, and timely data collection.

### 14.1 Statistical and Analytical Plans

The statistical analysis plan (SAP) will provide additional details on the planned statistical analysis and will be finalized prior to database lock. Unless otherwise stated, all analyses will be performed using SAS<sup>®</sup>.

### 14.1.1 Interim Analyses

Accruing study data will be summarized periodically for review by BioMarin. All summaries will be descriptive. Early stopping will be considered on the basis of safety only and will be based on clinical judgment; no inferential stopping rules will be employed.

## 14.2 Primary Efficacy Analysis

Because practical and ethical concerns preclude contemporaneous or untreated control subjects, CLN2 disease motor and language rating scale scores will be compared with historical data from existing CLN2 disease registries, as specified in the SAP.

### 14.3 Secondary Efficacy Analysis

The following parameters will be evaluated using descriptive statistics as outlined in the SAP:

 Various representations of brain volumes, as determined by MRI, will be summarized.

## 14.4 Exploratory Analyses

The following parameters will be evaluated, as specified in the SAP:

- Quality of life questionnaires
- Relationships among safety, immunogenicity and efficacy
- Denver II Developmental scale
- CSF/ blood biomarkers
- EEG, standard awake
- Preferential Looking Test; Optional Lea Vision Test or E Hook (or Tumbling E)
   Vision Test



Optical coherence tomography

# 14.5 Immunogenicity Analysis

Immunogenicity tests will be performed using validated immunogenicity assays on serum and CSF samples. Samples of CSF and serum will be collected for anti-BMN 190 TAb and NAb testing, as detailed in **Table 9.1.1**. Collection must precede study drug infusion when collected for routine immunogenicity assessments. Baseline blood (serum) samples will be collected at the Study Completion visit in Study 190-201 to obtain a baseline TAb and NAb, every 12 weeks thereafter (Q12W), at the Study Completion or Early Termination visit, at the Device Safety Follow-Up visit, and at the Safety Follow-Up visit. CSF samples will be collected for anti-BMN 190 TAb and NAb testing at the Study Completion visit in Study 190-201 and every 12 weeks thereafter (Q12W). Serum and CSF NAb will be tested at Study Completion Visit in Study 190-201 and at subsequent time points when serum and CSF TAb are positive, respectively. No CSF immunogenicity assessments will be performed at either of the safety follow-up visits.

Incidence and titer summary statistics will be provided for serum and CSF TAb and NAb in table format and will include mean, median, standard deviation, and minimum/maximum titer values at each study visit. Potential impact of anti-drug antibodies on efficacy and safety will be explored.

In the event of a suspected anaphylactic reaction, serious hypersensitivity event, or severe hypersensitivity (defined as a hypersensitivity event of Grade 3 or higher), blood samples to assess C4, serum tryptase, and total IgE will be collected within 1 hour of the event and tested; a blood sample to assess drug-specific IgE will be collected no sooner than 8 hours after the event (or before the next infusion). Potential associations between IgE positivity and hypersensitivity adverse events will be analyzed.

#### 14.6 Safety Analysis

All AEs will be coded by BioMarin using the current version of MedDRA to assign system organ class and preferred term classification to events and diseases, based on the original terms entered on the eCRF. The incidence of AEs will be summarized by system organ class, preferred term, relationship to study treatment, and severity for each dosing group.

Concomitant medications will be coded using World Health Organization Drug and summarized.



Clinical laboratory data will be summarized in terms of observed values and changes from Baseline. Lab data will also be summarized relative to categorical reference ranges (e.g., lab normal ranges and/or CTCAE grade).

Vital signs will be summarized in terms of observed values and changes from Baseline.

Results from continuous ECG monitoring (3- or 5-lead) and serial 12-lead ECGs will be descriptively summarized in terms of overall interpretation and abnormal findings. ECGs (12-lead) will be summarized in terms of investigator overall interpretation, abnormal findings, and quantitative intervals (QTcF, etc.).

# 14.7 Determination of Sample Size

The sample size will be determined by the number of subjects who complete Study 190-201 and decide to roll into Study 190-202. Up to 23 subjects are projected to enroll into Study 190-202.

## 14.8 Changes in the Conduct of the Study or Planned Analyses

Only BioMarin may modify the protocol. Any change in study conduct considered necessary by the investigator will be made only after consultation with BioMarin, who will then issue a formal protocol amendment to implement the change. The only exception is when an investigator considers a subject's safety compromised without immediate action. In these circumstances, immediate approval of the chairman of the IRB/IEC/REB must be sought, and the Investigator should inform BioMarin and the full IRB/IEC/REB within two (2) working days after the emergency occurs.

With the exception of minor administrative or typographical changes, the IRB/IEC/REB must review and approve all protocol amendments. Protocol amendments that have an impact on subject risk or the study objectives, or require revision of the ICF, must receive approval from the IRB/IEC/REB prior to their implementation.

When a protocol amendment substantially alters the study design or the potential risks or burden to subjects, the ICF will be amended and approved by BioMarin and the IRB/IEC/REB, and all active subjects must again provide informed consent.

Note: If discrepancies exist between the text of the statistical analysis as planned in the protocol and the final SAP, a protocol amendment will not be issued and the SAP will prevail.


|----------|---------------------|---------|
|----------|---------------------|---------|

# 15 DATA MONITORING COMMITTEE

No Data Monitoring Committee will be used for this study.



### 16 COMPENSATION, INSURANCE AND INDEMNITY

There will be no monetary compensation provided to subjects for their participation in this study. BioMarin is responsible for all study participation expenses, including tests, procedures, and treatments. In addition, BioMarin may reimburse the cost of travel for study-related visits after ethics committee approval. BioMarin will not pay for any hospitalization, tests, or treatments for medical problems not part of this protocol regardless of their relationship to the subject's disease. Costs associated with hospitalization, tests, and treatments should be billed and collected in the way that such costs would be customarily billed and collected

The investigator should contact BioMarin immediately upon notification that a study subject has an injury related to the study treatment or to the procedures or assessments performed as part of the study. Any subject who experiences a study-related injury should be instructed by the investigator to seek medical treatment at a pre-specified medical institution (if possible) or at the closest medical treatment facility (if necessary). The subject should be given the contact information if they require further information about or assistance with treatment for study-related injuries. The treating physician should bill the subject's health insurance company or other third party payer for the cost of this medical treatment. If the subject has followed the investigator's instructions, BioMarin will pay for reasonable and necessary medical services to treat the injuries caused by the study treatment or study assessments or procedures if these costs are not covered by health insurance or another third party that customarily would pay these costs. In some jurisdictions, BioMarin is obligated by law to pay for study-related injuries without prior recourse to third party payer billing. If this is the case, BioMarin will comply.



#### 17 CASE REPORT FORMS AND SOURCE DOCUMENTS

Electronic Case Report Forms (eCRFs) will be provided for each subject. eCRFs must be completed using a validated web-based application. Study site personnel or designee will be trained to enter the clinical data onto the eCRFs from source documentation using the web-based application. Unless explicitly allowed in the eCRF instructions, blank data fields are not acceptable.

The investigator must review and electronically sign the completed eCRF casebook to verify its accuracy.

In the event of an entry error, or if new information becomes available, the value will be corrected by deselecting the erroneous response and then selecting or entering the factual response. In compliance with US 21 CFR Part 11, the web-based eCRF system will require the personnel making the correction to enter a reason for changing the value.

The documented audit trail will include the reason for the change, the original value, the new value, the time of the correction, and the identity of the operator.

BioMarin policy is that study data on the eCRFs must be verifiable to source data, which necessitates access to all original recordings, laboratory reports, and subject records. In addition, all source data should be attributable (signed and dated). The investigator must, therefore, agree to allow direct access to all source data. Subjects (or legally authorized representative) must also allow access to their medical records. Subjects will be informed of the necessity for such access and will confirm their agreement with this when providing informed consent. If an investigator or institution refuses to allow access to subject records because of confidentiality, arrangements must be made to allow an "interview" style of data verification.

A BioMarin CRA (or designee) will compare eCRFs with original source documents at the study site and evaluate eCRFs for completeness and accuracy before designating them as "source data verified." If an error is discovered at any time or a clarification is needed, the CRA (or designee) will create an electronic query on the associated field. Study site personnel will then answer the query by either correcting the data or responding to the query. The CRA will then review the response and determine either to close the query or re-query the site if the response does not fully address the question. This process is repeated until all open queries have been answered and closed.

Before a subject eCRF casebook can be locked, data fields must be source data verified and all queries closed. Refer to the Study Monitoring Plan for details on which fields must be




source data verified. The investigator will then electronically sign the casebook, specifying that the information on the eCRFs is accurate and complete. The Data Manager (or designee) will then set the status of the forms, visits, and entire casebook to Locked. As part of site close-out activities, an electronic copy of each site's casebooks will be copied to a compact disc or digital versatile disc (DVD) and sent to each study site for retention with other study documents.



# 18 STUDY MONITORING AND AUDITING

Qualified individuals designated by BioMarin will monitor all aspects of the study according to GCP and standard operating procedures for compliance with applicable government regulations. The investigator agrees to allow these monitors direct access to the clinical supplies, dispensing, and storage areas and to the clinical files, including original medical records, of the study subjects, and, if requested, agrees to assist the monitors. The investigator and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by BioMarin or its designees.

Members of BioMarin GCP Compliance Department (or designee) may conduct an audit of a clinical site at any time before, during, or after completion of the study. The investigator will be informed if an audit is to take place and advised as to the scope of the audit. Representatives of the FDA or other regulatory agencies may also conduct an audit of the study. If informed of such an inspection, the investigator should notify BioMarin immediately. The investigator will ensure that auditors have access to clinical supplies, study site facilities, original source documentation, and all study files.



#### 19 RETENTION OF RECORDS

The investigator must retain all study records required by BioMarin and by the applicable regulations in a secure and safe facility. The investigator must consult a BioMarin representative before disposal of any study records, and must notify BioMarin of any change in the location, disposition, or custody of study files. The investigator and/or institution must take measures to prevent accidental or premature destruction of essential documents, that is, documents that individually and collectively permit evaluation of the conduct of a study and the quality of data produced, including paper copies of study records (e.g., subject charts) as well as any original source documents that are electronic as required by applicable regulatory requirements.

All study records must be retained for at least 2 years after the last approval of a marketing application in the US or an ICH region and until (1) there are no pending or contemplated marketing applications in the US or an ICH region or (2) at least 2 years have elapsed since the formal discontinuation of clinical development of the study drug. The investigator and/or institution should retain subject identifiers for at least 15 years after completion or discontinuation of the study. Subject files and other source data must be kept for the maximum period of time permitted by the hospital, institution, or private practice but not less than 15 years. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by a BioMarin agreement. BioMarin must be notified and will assist with retention should investigator and/or institution be unable to continue maintenance of subject files for the full 15 years. It is the responsibility of BioMarin to inform the investigator and/or institution when these documents no longer need to be retained.



# 20 USE OF INFORMATION AND PUBLICATION

BioMarin recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between BioMarin and the Investigator/Institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org/about-icmje/faqs/icmje-recommendations/) and good publication practices (GPP).



#### 21 REFERENCES

Arkin, LM, Sondhi, D, Worgall, S, Suh, LH et al. Confronting the issues of therapeutic misconception, enrollment decisions, and personal motives in genetic medicine-based clinical research studies for fatal disorders. Hum Gene Ther 16[9], 1028-1036. 2005.

Awano, T, Katz, ML, O'Brien, DP, Sohar, I et al. A frame shift mutation in canine TPP1 (the ortholog of human CLN2) in a juvenile Dachshund with neuronal ceroid lipofuscinosis. Mol Genet Metab 89[3], 254-260. 2006.

Brooks, R. EuroQol: the current state of play. Health Policy 37[1], 53-72. 1996.

Chang, M. CLN2. The Neuronal Ceroid Lipofuscinoses. New York: Oxford Univ Press, 2011: 80-109.

Crystal, RG, Sondhi, D, Hackett, NR, Kaminsky, SM et al. Clinical protocol. Administration of a replication-deficient adeno-associated virus gene transfer vector expressing the human CLN2 cDNA to the brain of children with late infantile neuronal ceroid lipofuscinosis. Hum Gene Ther 15[11], 1131-1154. 2004.

Dierenfeld, AD, McEntee, MF, Vogler, CA, Vite, CH et al. Replacing the enzyme alpha-Liduronidase at birth ameliorates symptoms in the brain and periphery of dogs with mucopolysaccharidosis type I. Sci Transl Med 2[60], 60ra89. 2010.

Dyke, JP, Sondhi, D, Voss, HU, Shungu, DC et al. Assessment of Disease Severity in Late Infantile Neuronal Ceroid Lipofuscinosis Using Multiparametric MR Imaging. AJNR Am J Neuroradiol. 2012.

Giedd, JN, Snell, JW, Lange, N, Rajapakse, JC et al. Quantitative magnetic resonance imaging of human brain development: ages 4-18. Cereb Cortex 6[4], 551-560. 1996.

Karavelis A, Foroglou G, Selviaridis P et al. Intraventricular administration of morphine for control for intractable cancer pain in 90 patients. Neurosurgery 39[1], 57-62. 1996.

Katz ML, Coates JR, Sibigtroth CM, Taylor JD et al. Enzyme replacement therapy attenuates disease progression in a canine model of late-infantile neuronal ceroid lipofuscinosis (CLN2 disease). J Neurosci Res 92[11], 1591-1598. 2014.

Kronenberg MF, Laimer I, Rifici C et al. Epileptic seizure associated with intracerebroventricular and intrathecal morphine bolus. Pain 75[2], 383-387. 1998.

Kurachi, Y, Oka, A, Mizuguchi, M, Ohkoshi, Y et al. Rapid immunologic diagnosis of classic late infantile neuronal ceroid lipofuscinosis. Neurology 54[8], 1676-1680. 2000.

Lishner M, Perrin RG, Feld R et al. Complications Associated with Ommaya Reservoirs in Patients with Cancer: The Princess Margaret Hospital Experience and a Review of the Literature. Arch Intern Med 150[1], 173-176. 1990.



Msall, M. Measuring Functional Skills in Preschool Children at Risk for Neurodevelopmental Disabilities. Ment. Retard. Dev. Disabil. Res. Rev. 11, 263-273. 2005.

Seitz, D, Grodd, W, Schwab, A, Seeger, U et al. MR imaging and localized proton MR spectroscopy in late infantile neuronal ceroid lipofuscinosis. AJNR Am J Neuroradiol 19[7], 1373-1377. 1998.

Sleat, DE, El-Banna, M, Sohar, I, Kim, KH et al. Residual levels of tripeptidyl-peptidase I activity dramatically ameliorate disease in late-infantile neuronal ceroid lipofuscinosis. Mol Genet Metab. 2008.

Sleat, DE, Wiseman, JA, El-Banna, M, Kim, KH et al. A mouse model of classical late-infantile neuronal ceroid lipofuscinosis based on targeted disruption of the CLN2 gene results in a loss of tripeptidyl-peptidase I activity and progressive neurodegeneration. J Neurosci 24[41], 9117-9126. 2004.

Schulz, A, Ajayi, T, Specchio, N, de Los Reyes, E, et al. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med 2018; 378[20]:1898-1907.

Steinfeld, R, Heim, P, von Gregory, H, Meyer, K et al. Late infantile neuronal ceroid lipofuscinosis: quantitative description of the clinical course in patients with CLN2 mutations. Am J Med Genet 112[4], 347-354. 2002.

The EuroQol Group. EuroQol-a new facility for the measurement of health-related quality of life. Health Policy 16[3], 199-208. 1990.

Vuillemenot, BR, Katz, ML, Coates, JR, Kennedy, D et al. Intrathecal tripeptidyl-peptidase 1 reduces lysosomal storage in a canine model of late infantile neuronal ceroid lipofuscinosis. Mol Genet Metab 104[3], 325-337. 2011.

Vuillemenot, BR, Kennedy, D, Reed, RP, Boyd, RB, et al. Recombinant human tripeptidyl peptidase-1 infusion to the monkey CNS: safety, pharmacokinetics, and distribution. Toxicol Appl Pharmacol 277[1], 49-57. 2014.

Worgall, S, Kekatpure, MV, Heier, L, Ballon, D et al. Neurological deterioration in late infantile neuronal ceroid lipofuscinosis. Neurology 69[6], 521-535. 2007.

Worgall, S, Sondhi, D, Hackett, NR, Kosofsky, B et al. Treatment of late infantile neuronal ceroid lipofuscinosis by CNS administration of a serotype 2 adeno-associated virus expressing CLN2 cDNA. Hum Gene Ther 19[5], 463-474. 2008.

Xu, S, Wang, L, El-Banna, M, Sohar, I et al. Large-volume intrathecal enzyme delivery increases survival of a mouse model of late infantile neuronal ceroid lipofuscinosis. Mol Ther 19[10], 1842-1848, 2011.



#### 22 INVESTIGATOR RESPONSIBILITIES

# 22.1 Conduct of Study and Protection of Human Subjects

In accordance with FDA Form 1572, the Investigator will ensure that:

- He or she will conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.
- He or she will personally conduct or supervise the study.
- He or she will inform any potential subjects, or any persons used as controls, that the drugs are being used for investigational purposes and he or she will ensure that the requirements relating to obtaining informed consent in 21 CFR Part 50 and IRB review and approval in 21 CFR Part 56 are met.
- He or she will report to the sponsor adverse experiences that occur in the course of the investigation in accordance with 21 CFR 312.64.
- He or she has read and understands the information in the Investigator's Brochure, including potential risks and side effects of the drug.
- His or her staff and all persons who assist in the conduct of the study are informed about their obligations in meeting the above commitments.
- He or she will ensure that adequate and accurate records in accordance with 21 CFR 312.62 and to make those records available for inspection in accordance with 21 CFR 312.68
- He or she will ensure that the IRB/EC/REB complies with the requirements of 21 CFR Part 56, and other applicable regulations, and conducts initial and ongoing reviews and approvals of the study. He or she will also ensure that any change in research activity and all problems involving risks to human subjects or others are reported to the IRB/EC/REB. Additionally, he or she will not make any changes in the research without IRB/EC/REB approval, except where necessary to eliminate apparent immediate hazards to human subjects.
- He or she agrees to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements in 21 CFR Part 312.



### 23 SIGNATURE PAGE

**Protocol Title:** A Multicenter, Multinational, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 190 in Patients with CLN2 Disease

**Protocol Number:** 190-202

I have read the forgoing protocol and agree to conduct this study as outlined. I agree to conduct the study in compliance with all applicable regulations and guidelines, including E6 ICH, as stated in the protocol, and other information supplied to me.

| Investigator Signature | | Date |
|---|---|---|
| Printed name: | | |
| Accepted for the Sponsor: | DocuSigned by: PI Signer Name: PI Signing Reason: I approve this document Signing Time: 12/21/2018 3:28:03 PM PST CF6CF33D7AD74E5595998DB29C6C09E8 | |
| Medical Monitor Signature | | Date |

, MD

Sr. Medical Director, Rare Disease

Printed name: PI

|----------|---------------------|---------|
|----------|---------------------|---------|

# 24 APPENDICES

# Appendix 1: Adapted CLN2 Disease Rating Scale

| | Ham | burg LINCL Scale (Steinfeld, 2002),<br>adapted for multicenter use | | We | eill Cornell LINCL Scale (Dyke, 2012),<br>adapted for multicenter use |
|---|---|---|---|---|---|
| Motor / Gait | 3 | Grossly normal gait. No prominent ataxia, no pathol | logic falls | | |
| | 2 | Independent gait, as defined by ability to walk without support for 10 steps. Will have obvious instability, and may have interm falls. Requires external assistance to walk, or can crawl only. | | | |
| | 1 | | | | |
| | 0 | Can no longer walk or crawl. | | | |
| Language | 3 | Apparently normal language. Intelligible and grossly | y age-appropriat | e. No de | ecline noted yet. |
| | 2 | Language has become recognizably abnormal: some intelligible words, may form short sentences to convey concepts, reque needs. This score signifies a decline from a previous level of ability (from the individual maximum reached by the child). | | | |
| | 1 | Hardly understandable. Few intelligible words | | | |
| | 0 | No intelligible words or vocalizations | | | |
| Vision | 3 | Grossly normal. Appears to recognize multiple objects and reacts appropriately (reaches for a toy, etc.) | Myoclonus | 3 | No myoclonus, involuntary movements. Babinski not present |
| | 2 | Apparent difficulty seeing some objects. May be able to discern large objects, moving objects, but vision is clearly impaired. This score signifies a decline from a previous level of ability. | | 2 | One finding: (myoclonus) (chorea, dystonia, tremor, athetosis) (Babinski present) |
| | 1 | Reacts only to light | | 1 | Two findings: (myoclonus) (chorea, dystonia, tremor, athetosis) (Babinski present) |
| | 0 | No reaction to light | | 0 | Myoclonus, involuntary movements, and Babinski present |

|----------|---------------------|---------|
|----------|---------------------|---------|

| Hamburg LINCL Scale (Steinfeld, 2002),<br>adapted for multicenter use | | Weill Cornell LINCL Scale (Dyke, 2012), adapted for multicenter use | | | |
|---|---|---|---|---|---|
| Seizures (grand mal) | 3 | No seizures in 12-week period | Feeding | 3 | No swallowing dysfunction |
| | 2 | 1 to 2 seizures in 12-week period | | 2 | Mild swallowing dysfunction but tolerates most food / drinks |
| | 1 | 3 seizures in 12-week period (1 per 4 weeks) | | 1 | Moderate swallowing dysfunction: difficulty with many foods |
| | 0 | > 3 seizures in 12-week period (> 1 per 4 weeks) | | 0 | Gastrostomy tube dependent |

|----------|---------------------|---------|
|----------|---------------------|---------|

## 25 PROTOCOL AMENDMENT TEXT REVISIONS

The following is a summary of significant protocol revisions; added text is <u>underlined</u> and deleted text is <u>struck</u>. Additional administrative changes have been made for consistency and clarity throughout this amendment and are reflected in the protocol body.

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Synopsis/Study Design<br>9.1/ Study Design and Plan | Patients will complete safety and efficacy assessments including CSF surveillance labs every 2 weeks, CLN2 disease scales every 8 weeks, and physical examination, clinical laboratory assessments, visual acuity tests, and immunogenicity tests every 12 weeks. MRI_MRI will be performed every 24 weeks. In addition, quality of life measures, OCT, EEG, developmental milestones (Denver II), will be completed, and blood and CSF samples for evaluating disease-related biomarkers will be collected every 24 weeks. Complete physical examination will be performed every 48 weeks. | 3, 6, 8 |
| Synopsis/Criteria for Evaluation | <ul> <li>electrocardiogram (ECG), 3- or 5-lead, 12-lead</li> <li>EEG, standard awake</li> <li>immunogenicity, includes anti-BMN 190 total antibodies (TAb) and neutralizing antibodies (Nab) in CSF; and TAb, NAb, and TAb titers and total IgE, and drug-specific IgE positivity in serum</li> </ul> | |
| | <ul> <li>Efficacy:</li> <li>CLN2 disease rating scales with videotaping</li> <li>Total cortical grey matter volume</li> <li>Quality of Life surveys</li> <li>Developmental assessments (exploratory)</li> <li>Disease-related biomarkers (exploratory)</li> <li>EEG, standard awake</li> <li>Assessments of visual acuity</li> <li>Optical coherence tomography</li> <li>Neurological Exam</li> </ul> | 1, 3, 6 |

|----------|---------------------|---------|
|----------|---------------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| Synopsis/ Statistical | Immunogenicity: anti-BMN 190 total antibodies (TAb) and neutralizing antibodies (NAab) in CSF; and TAb, NAb, total IgE, and drug-specific and anti-BMN 190-IgE in serum. Safety assessments include adverse events, clinical laboratory results, vital signs, ECGs, EEGs, and immunogenicity. | 3 |
| Methods | Efficacy data include CLN2 assessments and MRI measurements of brain volumes. | <u>.</u> |
| 6/ Investigators and Study<br>Administrative Structure | Assessment of immunogenicity and disease-related biomarkers will be conducted by BioMarin. Clinical laboratory evaluations will be performed by local study site laboratories. Central laboratories will be used to evaluate TPP1 enzyme activity, magnetic resonance imaging (MRI) scans, and electroencephalograms (EEGs). Additional details will be provided in the corresponding Study Laboratory Manual. | 3, 4 |
| 7.2/ Previous Clinical Studies | BMN 190 has been studied in human The only previous-clinical trials 190-experience with this investigational product is the BMN 190-201 and 190-202. Study 190-201 was trial, a 48 -week, international, multicenter phase 1/2 open-label dose-escalation study designed to assess the safety and efficacy of BMN 190 administered to patients with mild to moderate CLN2 disease by direct intracerebroventricular infusion to the CNS; Study 190-202 is the open-label extension of 190-201. This study enrolled 24 subjects at least 3 years of age (mean 4.3 years, range 3.8 years) with a two domain CLN2 disease score of 3 - 6 on motor and language domains of the Hamburg Scale (mean total score 3.7, SD=0.95), with a score of at least 1 in each of these two domains. Fifteen subjects (63%) were female and 9 (38%) subjects were male. These subjects were enrolled in 3 cohorts which received escalating doses of BMN 190 and a final cohort who received stable dose of drug. The first 3-subject cohort received 300 mg ow infusions, the second 3 subject cohort received 100 mg qow infusions and the third 4 subject cohort received 300 mg infusions of BMN 190. A final 14 subject cohort received a stable dose of 300 mg of BMN 190 during their participation in the study. A single patient withdrew consent from the study (subject 1287-1007) after ICV reservoir placement and a single infusion because of inability to comply with study procedures. Therefore, the efficacy population comprised 23 of the 24 subjects enrolled into Study 190-201. These studies evaluated the safety, tolerability and efficacy of BMN 190 given as an infusion of 300 mg every 14 days given directly to the CNS using a permanently implanted intracerebroventricular (ICV) access device. A total of 24 patients with screening CLN2 motor-language scores ≥ 3 (0 to 6 point scale) and age ≥ 3 were enrolled into the 190-201 study. All completers without predefined stopping criteria were qualified to enroll into the long term | 12 |

|----------|---------------------|---------|
|----------|---------------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | All patients had successful surgical implantation of ICV access devices, with device complication rates consistent | |
| | with what has been observed in the published literature. | |
| | Interim results of the completed 48-week open-label study (190-201) and the ongoing extension study (190-202) have | |
| | been published (Schulz, 2018, N Engl J Med). The primary outcome measure was the time until a 2-point decline in | |
| | the score on the motor and language domains of the CLN2 Clinical Rating Scale (which ranges from 0 to 6, with 0 | |
| | representing no function and 3 representing normal function in each of the two domains), which was compared with | |
| | the time until a 2-point decline in 42 historical controls. Additionally, rate of decline in motor–language score was | |
| | compared between the two groups using data from baseline to the last assessment with a score of more than 0, divided | |
| | by the length of follow-up (in units of 48 weeks). | |
| | Twenty-four subjects were enrolled in Study 190-201/190-202, 23 of whom constituted the efficacy population. | |
| | Interim efficacy results demonstrated a statistically significant and durable treatment effect in attenuating disease | |
| | progression as measured by CLN2 scores and in comparison to natural history. Of the 24 patients enrolled into | |
| | Study190-201, all but 2 subjects were in the active loss of function phase of the disease characterized by both notable | |
| | disease burden and decline by a median value of 2 points per 48 weeks. In the 23 subjects who received BMN 190 for | |
| | at least 96 weeks in Study 190-201/190-202, the median time until a 2-point decline in the motor-language score was | |
| | not reached and was 345 days for historical controls. The mean (SD) unadjusted rate of decline in the motor–language | |
| | score per 48-week period was 0.27 (0.35) points in treated subjects and 2.12 (0.98) points in 42 historical controls | |
| | (mean difference, 1.85; P < 0.001). Common AEs included convulsions, pyrexia, vomiting, hypersensitivity reactions, | |
| | and failure of the intraventricular device. In 2 subjects, infections developed in the intraventricular device that was | |
| | used to administer the infusion, which required antibiotic treatment and device replacement. | |
| | PK analysis of ICV-delivered BMN 190 demonstrates concentrations and exposures that are three orders of | |
| | magnitude greater in the CSF than in the plasma. | |
| | No association was found between ADA, including drug-specific IgE positivity, and incidence or severity of | |
| | hypersensitivity adverse events. | |
| | Taken together, the response in the treated group is significant when compared to the loss of function predicted by | |
| | natural history studies. The conclusions of treatment effect are constant across all analysis methodologies and | |
| | sensitivity analyses. Most patients (87%) experience neurodegenerative stabilization, in which active decline in | |
| | function is either halted (57%), has an early single point decline with no subsequent loss (22%) or actually improves | |
| | function on treatment (9%). | |
| | In conclusion, BMN 190 via ICV infusion is generally safe and well tolerated. BMN 190 treatment demonstrated a | |
| | durable and clinically meaningful therapeutic effect on attenuating disease progression compared to natural history. | |

|----------|---------------------|---------|
|----------|---------------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | All doses of BMN 190 administered were generally well tolerated and there were no early terminations due to adverse events in this study. The occurrence and severity of adverse events, particularly those related to hypersensitivity, did not appear to be associated with higher doses of BMN 190. Results from the 190 201 study demonstrated a substantial improvement of the rate of clinical progression in children treated with BMN 190 compared with untreated historical controls. Further, in those children who had received at least 48 weeks of BMN 190 dosing, clinical scores stabilized, in contrast to matched historical untreated controls in which decline was rapid and profound in the majority of matches. | |
| 7.4/ Summary of Risks and<br>Benefits | Nonclinical toxicity No findings in any of the six nonclinical studies have not identified drug indicate adverse BMN 190-related adverse effects associated on cardiovascular or central nervous systems. Electrocardiogram (ECG) analysis in cynomolgus monkeys revealed no changes in ECG waveform or heart rate after a single ICV infusion during the time of BMN 190 exposure in the CSF and plasma. | |
| | Although a stand alone CNS safety pharmacology study was not conducted, monthly neurologic and clinical examinations of dachshunds administered BMN 190 (4 or 16 mg) for 9 months in a repeated infusion study revealed no clinical CNS signs in dachshunds attributable to BMN 190. CNS signs known from historical control data to be due to disease progression in this model (ataxia, tremor, myoclonus, proprioceptive deficits, and visual decline) were observed in treated and untreated TPP1 null dachshunds (Awano, 2006, Mol.Genet.Metab), (Katz, 2014, J.Neurosci.Res.). Furthermore, onset of disease related neurologic signs was delayed 3.5 to 11 weeks following 4 mg BMN 190 and 10 to 28 weeks following 16 mg BMN 190, compared with chronic vehicle treated controls. | 12 |
| | Given the lack of BMN 190-related safety concerns of these studies, the specific mechanism of BMN 190 action, and that nearly all (- 99%) BMN 190 remains in the CNS after ICV administration of BMN 190 to healthy or CLN2 animal models disease, untoward systemic safety effects are unlikely in human. BMN 190 has been studied in 24 patients in 5 clinical sites for Studies 190-201 and 190-202. The current clinical experience in human clinical trials demonstrates an acceptable benefit-risk profile to both the placement and chronic use of ICV access devices, and to infusion of BMN 190 at 300 mg every 14 days as demonstrated by interim efficacy and safety results summarized in Section 7.2. Furthermore, efficacy analysis of Study 190 201 showed an | |

BIOMARIN" 190-202 Amendment 6 Page 97

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | attenuation of the decline in motor language scores on the Hamburg CLN2 clinical rating scale, which when matched to members of the Hamburg natural history cohort by baseline score, age and genotype showed significant treatment benefit for BMN 190. Of the 24 patients enrolled into Study190 201, all but 2 patients were in the active loss of function phase of the disease characterized by both notable disease burden and decline by a median value of 2 points each year (0 to 6 point scale). Treatment during this stage protected further decline in the disease. | |
| | The efficacy objective of this study is to prevent patients from entering into the active rapid loss of function phase of the disease, or to attenuate further progression of disease. Monitoring and evaluation of specific adverse events of hypersensitivity reactions and device-related complications are discussed in Sections 7.4.1 and 7.4.2. Given the severity of disease, clinical and nonclinical support of possible efficacy, the overall risks and benefits support this protocol. | |
| 7.4.2/ Risk of ICV Devices and Drug Administration | New text: Material degradation of the ICV device reservoir has occurred after approximately 105 perforations of the ICV device in benchtop testing, and has been observed in clinical trials with approximately 4 years of BMN 190 administration. Access device replacement should be considered prior to 4 years of regular administration of BMN 190; with the decision made on an individual subject level based on the medical judgment of the Investigator. | 9 |
| Table 9.1.1/SOE | Changes to the SOE table and footnotes have been made to be consistent with changes made elsewhere in the protocol. | |
| 9.3.3.1/ Stopping Criteria | Subjects with a score of 0 on the combined motor and language components of the Hamburg CLN2 rating scale at two consecutive visits without any change will be removed discontinued from treatment the study. | 10 |
| 9.3.5/ Duration of Subject<br>Participation | A Safety Follow-Up visit will be conducted 6 months after the final BMN 190 infusion. The Safety Follow-Up visit will be waived for subjects who receive study drug in another BioMarin-sponsored study or registry within this 6-month period (refer to Section 10.1 and Section 10.2 for AE and SAE reporting instructions). For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug. | 2 |

190-202 Amendment 6

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 9.4.4.1/ Safety Monitoring 9.7.5.2/ Device Malfunction 10.3/ Adverse Events of Special Interest 12.3/ Study Completion or Early Termination Visit | All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, defined in the protocol) should also be returned. | 11 |
| 9.4.7/ Blinding | Oversight of EEG evaluation will be performed by an independent epileptologist at a central facility. The interpreting epileptologists and software analysis will be blinded to subject and time on study. All subject-identifying information will be redacted before endpoints are assessed. | 3, 4 |
| 9.7 /Efficacy and Safety<br>Variables | Although this study is designed to assess safety and tolerability primarily, efficacy will be assessed by impact on disease-specific clinical rating scales. Secondary variables include MRI is being assessed as a secondary efficacy variable, and effect Effect on quality of life (QoL), developmental milestones,).—Disease-related biomarkers, EEG, visual acuity, and optical coherence tomography (OCT) and developmental milestones will also be explored. | 3, 6 |
| 9.7.3.1/ Quality of Life<br>Testing | Quality of life will be assessed using 23 different instruments: the PedsQL <sup>TM</sup> Measurement Model for Pediatric Quality of Life Inventory (PedsQL)), the EuroQol Health Status EQ 5D 5L Instrument, and the CLN2-specific questionnaire. | 7 |
| 9.7.2.2.2/ EuroQol Health<br>Status EQ-5D-5L<br>Instrument | The EQ 5D 5L instrument is a self-reported questionnaire designed to measure general health status (The EuroQol Group, 1990, Health Policy), (Brooks, 1996, Health Policy). The EQ-5D-5L is composed of 2 parts: a descriptive system that assesses 5 levels of perceived problems (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) in 5 dimensions and the EQ visual analogue scale (EQ VAS) assessment for overall health. | 7 |

|----------|---------------------|---------|
|----------|---------------------|---------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 9.7.3.4/<br>Electroencephalogram | Moved: A standard awake EEG will be recorded within 2 days before each infusion as indicated in Table 9.1.1. If a clinically significant abnormality is noted, the investigator or designee will evaluate whether study enrollment or continuation is appropriate; a clinically significant abnormality will be recorded under Medical History during Week 1 and as an AE thereafter. Evaluation will be done both locally and by a centralized vendor. | 3, 4 |
| 9.7.3.5/ Assessments of Visual Acuity | The Preferential Looking Test (PLT) is a method of assessing visual acuity in infants and children with limited cognitive function. The PLT assesses the acuity of children who are unable to identify pictures, shapes, or letters, and is particularly useful in children with physical and/or mental disabilities. The principle of the test is that a young child will choose to look towards an interesting visual stimulus ("target") rather than a plain stimulus. The child is presented with two stimulus fields, one with stripes and the other with a homogeneous gray area of the same average luminance as the striped field. The location of the stripes is randomly alternated. Typically, infants and children will look at the more interesting stripes (if they can detect them) rather than at the blank field. Teller, Keeler, and LEA Grating Acuity Cards have been standardized to assess grating (resolution) visual acuity in infants and nonverbal children using the principles of Preferential Looking. Other standardized versions of the LEA Test System use symbols or numbers to assess visual acuity in children who do not know how to read the letters of the alphabet that are typically used in an eye chart, but require higher cognitive function than PLT. The symbols are likely to be more useful in the CLN2 patient population. Similarly, the E-Hook or Tumbling E chart has been standardized to use rows of the letter "E" in various orientations. The patient is asked to point to where the limbs of the E are pointing "up, down, left or right." Depending on how far down the chart the patient can "read", his or her visual acuity is quantified. All subjects will perform PLT. Use of standardized Teller, Keeler, or LEA Grating Cards to perform PLT are all acceptable based on institutional standards and availability of personnel experienced in performing the assessments. The choice of testing materials should be consistent for all patients at each investigational site. In addition, for those children who retain the cognitive function to adhere | 6 |

|----------|---------------------|----------|--|
|----------|---------------------|----------|--|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | for higher functioning children (eg, LEA symbol or Tumbling E) should be made based on availability of experienced and qualified personnel to perform the assessment and should remain consistent throughout the study. Whenever | |
| | possible, all tests of visual acuity should be performed by the same tester. The tests of visual acuity may be done either before or after drug infusion based on logistical considerations and ease for the subject and study personnel. However, the timing should remain consistent for all subsequent assessments. Patients must be alert and not influenced by any sedating medications. | |
| 9.7.3.6/ Optical Coherence<br>Tomography | Optical coherence tomography (OCT) is a non-invasive imaging test that uses light waves to take cross-sectional pictures of the retina's layers in order to measure their thickness. These measurements can aid in early detection and treatment for retinal diseases. OCT will be performed locally and should precede infusions. In order to limit the need for sedation to perform this assessment, measurement should be obtained while the subject is also under sedation for MRI acquisition. OCT images will be collected by BioMarin, to be assessed by BioMarin personnel or designees. | 6 |
| 9.7.4/Immunogenicity | Immunogenicity tests will be performed using validated immunogenicity assays on serum and CSF samples. Samples of blood (serum) will be collected for anti-BMN 190 TAb testing, and Samples of CSF and serum will be collected for anti-BMN 190 TAb and NAb testing, as detailed in Table 9.1.1. Collection must precede study drug infusion when collected for routine immunogenicity assessments. Baseline blood (serum) samples will be collected at the Study Completion visit in Study 190-201 to obtain a baseline TAb and NAb, every 12 weeks thereafter (Q12W), at the Study Completion or Early Termination visit, at the Device Safety Follow-Up visit, and at the Safety Follow-Up visit. CSF samples will be collected for anti-BMN 190 TAb and NAb testing at the Study Completion visit in Study 190-201 and every 12 weeks thereafter (Q12W). Serum and CSF NAb samples will be tested at Study Completion Visit in Study 190-201 and at subsequent time pointsonly when serum and the corresponding-CSF TAb are sample | 1 |

|----------|---------------------|----------|
|----------|---------------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | tests-positive, respectively. No CSF immunogenicity assessments will be performed at either of the safety follow-up visits. | |
| 9.7.6.2/ Physical<br>Examination | A <u>complete</u> physical examination will be performed as indicated in Table 9.1.1. A complete examination will include general appearance (head, eyes, ears, nose, and throat), cardiovascular, dermatologic, lymphatic, respiratory, gastrointestinal, genitourinary, musculoskeletal, <u>and</u> neurologic systems (level of consciousness, speech, language, cranial nerves, motor strength, motor tone, abnormal movements, reflexes, upper extremity sensation, lower extremity sensations, gait, Romberg, nystagmus, and coordination).), and body weight and height. Results of the neurologic examination may also be used to assess the efficacy of BMN 190. | |
| | A <u>brief</u> physical examination will be performed otherwise, as indicated in Table 9.1.1. A brief examination will include general appearance, cardiovascular, respiratory, neurologic, and gastrointestinal assessments. | |
| | Body weight and height assessments should be performed at the timepoints indicated in Table 9.1.1. | |
| | Use of an ICV reservoir device for intracerebroventricular drug administration requires that patients be monitored throughout the study for potential infections (high temperature, cough, rash, headache, mental status changes, swelling or drainage in the incision area) and signs of ICV reservoir leakage or failure (swelling of skin around reservoir site, difficulty with CSF extraction, erythema of the scalp, bulging of reservoir device, or extravasation of fluid on infusion). | 8, 9, 11 |
| | The investigator will evaluate the patency, location, and skin integrity of the reservoir at each study drug administration. The investigator will check for scalp edema, erythema or skin breakdown at the site of the reservoir prior to infusion. Patency will be assessed during pre-infusion sampling and again at the time of infusion. Difficulty in obtaining the required volume of CSF necessary for pre-infusion samples or signs of ICV reservoir leakage (swelling of skin around reservoir site, erythema of the scalp, bulging of reservoir device, or extravasation of fluid) will prompt further evaluation of the reservoir for failure prior to continuing with infusion. Additional surgical consultation including surgery may be required to revise or replace the device. Material degradation of the ICV device reservoir has occurred after approximately 105 perforations of the ICV device in benchtop testing, and has | |

|----------|---------------------|----------|
|----------|---------------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 10.1/Adverse Events | been observed in clinical trials with approximately 4 years of BMN 190 administration. Access device replacement should be considered prior to 4 years of regular administration of BMN 190; with the decision made on an individual subject level based on the medical judgment of the Investigator. All removed or replaced implantable ICV devices must be returned to BioMarin in order to evaluate the material integrity of the reservoir, and all other devices (as described in the Pharmacy Manual) except for infusion pumps, defined in the protocol) should also be returned. All AEs/ SAEs/ adverse events of special interest (AEOSIs) / pregnancies will be recorded starting after the first dose of study drug in Study 190-202. Reporting of AEs/SAEs / AEOSIs/ pregnancies will continue until 6 months after either the last administration of study drug or the Early Termination visit. The 6-month Safety Follow-Up Visit will be waived for subjects who begin receiving study drug in another BioMarin-sponsored study or registry within this 6-month period. For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the time of the last dose or new events related to study drug. For this study, a medical device is defined as the infusion pump and all contact parts components required for infusion (reservoir and catheter, needles, infusion line with filter, extension sets, and syringes) intended to be used for administration of BMN 190. Adverse events assessed by the investigator as related to the device, including malfunction, injury, or medication error, will be entered into the device AE/SAE eCRF and the device report form and reported to BioMarin Pharmacovigilance (BPV) within 24 hours by entering the event information via EDC and completing the study specific device report form(s). Prophylactic replacement of the ICV must be reporting period for device-related | 2, 9 |
| 10.2/ Serious Adverse<br>Events | The reporting period for SAEs begins after the first dose of study drug in Study 190-202 and continues until 6 months after either the last administration of study drug or the Early Termination visit. The 6-month Safety Follow-Up Visit will be waived for subjects who begin receiving study drug in another BioMarin-sponsored study or registry within this 6-month period. Refer to Section 10.1 for additional information regarding SAE reporting for these subjects. For subjects who do not participate in an extension study or registry after the last dose of study drug, the 4-week device | 2 |

|----------|---------------------|----------|
|----------|---------------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | safety follow-up visit and 6-month safety follow-up visit will capture information regarding ongoing events at the | |
| | time of the last dose or new events related to study drug. If a subject is discontinued from the study prematurely, SAEs will be recorded at the Early Termination visit. | |
| 10.4.8/ Hospitalization,<br>Prolonged Hospitalization,<br>or Surgery | Perform a protocol-mandated procedure (excludes prophylactic ICV replacement) | 9 |
| 12.1/ Screening/ Baseline | The following procedures will be performed during the Screening Period: | |
| - | Informed consent/assent | |
| | Criteria for study entry | |
| | Pregnancy testing | 7 |
| | • EQ 5D 5L | |
| 12.2.3/ Every 12 Weeks | Every 12 weeks (± 3 days) (Weeks 13, 25, 37, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, 169, 181, 193, 205, 217, 229), the following procedures will be performed: • CSF/serum for immunogenicity | |
| | Complete physical examination | |
| | Visual acuity testing | |
| | All subjects will undergo Preferential Looking Testing every 12 weeks. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or E Hook (or Tumbling E) Vision Test should also be performed during the same assessment. Visual acuity testing can be performed either before or after the infusion (± 3 days), but should be performed at a time (relative to infusion) that can be repeated consistently between study visits. The subject must not be sedated at the time of visual acuity testing. | 6 |

190-202 Amendment 6

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 12.2.4/ Every 24 Weeks | Every 24 weeks (± 3 days) (Weeks 25, 49, 73, 97, 121, 145, 169, 193, 217), the following procedures will be performed: • Height and body weight assessment • CLN2 disease rating scales with videotaping • ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities) 30 (±5) minutes after infusion end • EEG, standard awake • MRI (±4-week window is allowed for this assessment and may be performed at the same time as a scheduled infusion) • CSF/ blood for disease-related biomarkers • Optical coherence tomography • CLN2-specific QoL questionnaire • PedsQL • EQ 5D 5L • Denver II Developmental Scale | 6, 7, 8 |
| 12.2.5/ Every 48 Weeks | The following procedures should be performed every 48 weeks during the study: • Complete physical examination | 8 |

190-202 Amendment 6

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 12.3/ Study Completion or<br>Early Termination Visit | The Study Completion visit will occur 2 weeks (± 3 days) after the last dose of BMN 190 (Week 239), or within 1 week of early study termination. At the Study Completion or Early Termination visit, the following procedures will be completed: | |
| | Hamburg and Weill Cornell CLN2 disease rating scales (Appendix 1) videotaped | |
| | ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities) | |
| | EEG (standard awake) | |
| | • MRI (±4-week window is allowed for this assessment and may be performed at the same time as a scheduled infusion) | |
| | CSF surveillance (cell count, protein, glucose, and culture) | |
| | CSF and blood for biomarker assays | |
| | CSF and serum for immunogenicity (TAb; NAb if TAb positive) | |
| | Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate) | 6, 7, 8, 13 |
| | Complete physical examination, including neurologic examination | |
| | Height, including neurological examination and body weight assessment | |
| | Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis) | |
| | • PedsQL | |
| | <u>Visual acuity testing</u> | |
| | <ul> <li>All subjects will undergo Preferential Looking Testing. In addition, for those children who retain the cognitive function to adhere to testing, the Lea Vision Test or E Hook (or Tumbling E) Vision Test should also be performed during the same assessment.</li> </ul> | |
| | Optical coherence tomography | |
| | ● EQ 5D 5L | |


| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | CLN2-specific QoL questionnaire | |
| | Denver II Developmental scale | |
| | Neurological examination | |
| | <ul> <li>AE assessment (investigator may collect additional blood samples for safety or immunogenicity testing for<br/>any AE of concern)</li> </ul> | |
| | Concomitant medication assessment | |
| 12.4/ Device Safety<br>Follow-Up Visit | Subjects will return to the study site 4 weeks (±3 days) after removal of the ICV access device, when the following procedures will be completed: | |
| | <u>CLN2 disease rating scales (videotaping not required)</u> | |
| | <ul> <li>Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate)</li> </ul> | |
| | <ul> <li>Brief physical examination (including close examination of the former device site to check for signs of<br/>infection, etc.)</li> </ul> | |
| | Neurological examination | |
| | Serum for immunogenicity (TAb) | 2, 5 |
| | Serum for total IgE, C4, and tryptase | |
| | Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis) | |
| | <ul> <li>AE assessment (investigator may collect additional blood samples or CSF by lumbar puncture for safety or<br/>immunogenicity testing for any AE of concern), including ongoing events at the time of the last dose or new<br/>events related to study drug.</li> </ul> | |
| | Concomitant medication assessment | |

190-202 Amendment 6

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| 12.5/ Safety Follow-Up | Subjects will return to the study site 6 months after the last study treatment, when the following procedures will be completed: | |
| | <u>CLN2 disease rating scales (videotaping not required)</u> | |
| | ECG (12-lead) (heart rate, rhythm, intervals, axis, conduction defects, and anatomic abnormalities) | |
| | EEG (standard awake) | |
| | Serum for immunogenicity (TAb) | |
| | • Serum for total IgE, C4, and tryptase | |
| | • Vital signs (SBP, DBP, heart rate, oral body temperature, and respiration rate) | 2, 5, 8 |
| | Complete physical examination | 2, 3, 6 |
| | Height and body weight assessment | |
| | Routine clinical laboratory tests (hematology, blood chemistry, and urinalysis) | |
| | <ul> <li>AE assessment (investigator may collect additional blood samples for safety or immunogenicity testing for<br/>any AE of concern), including ongoing events at the time of the last dose or new events related to study<br/>drug.</li> </ul> | |
| | Concomitant medication assessment | |
| 14.4/ Exploratory Analyses | The following parameters will be evaluated, as specified in the SAP: | |
| 1 7 7 | Quality of life questionnaires | |
| | Relationships among safety, immunogenicity and efficacy | 3, 6, 13 |
| | Denver II Developmental scale | |
| | <u>CSF/ blood biomarkers</u> | |

|----------|---------------------|----------|
|----------|---------------------|----------|

| Section | Revision | Rationale for<br>Change |
|---|---|---|
| | <ul> <li>EEG, standard awake</li> <li>Preferential Looking Test; Optional Lea Vision Test or E Hook (or Tumbling E) Vision Test</li> <li>Optical coherence tomography</li> </ul> | |
| 14.5/ Immunogenicity<br>Analysis | Immunogenicity tests will be performed using validated immunogenicity assays on serum and CSF samples. Samples of CSF and serum will be collected for anti-BMN 190 TAb and NAb testing, as detailed in Table 9.1.1. Collection must precede study drug infusion when collected for routine immunogenicity assessments. Baseline blood (serum) samples will be collected at the Study Completion visit in Study 190-201 to obtain a baseline TAb and NAb, every 12 weeks thereafter (Q12W), at the Study Completion or Early Termination visit, at the Device Safety Follow-Up visit, and at the Safety Follow-Up visit. CSF samples will be collected for anti-BMN 190 TAb and NAb testing at the Study Completion visit in Study 190-201 and every 12 weeks thereafter (Q12W). Serum and CSF NAb will be tested at Study Completion Visit in Study 190-201 and at subsequent time points when serum and CSF TAb are positive, respectively. No CSF immunogenicity assessments will be performed at either of the safety follow-up visits. Samples of blood (serum) will be collected for anti-BMN 190 TAb testing and samples of CSF will be collected for anti-BMN 190 TAb and NAb testing before the first infusion (i.e., at the completion of Study 190-201) and every 12 weeks thereafter or within one week of the Early Termination visit, CSF NAb samples collected prior to first infusion and will be tested at subsequent immunogenicity time points only when the CSF TAb is positive. Total IgE, C4, and tryptase samples will be collected prior to first infusion and within 1 hour of a hypersensitivity event. Collection must precede study drug infusion when collected for routine immunogenicity assessments. Incidence and titer summary statistics will be provided for serum TAb, CSF TAb, and CSF TAb and NAb in table format and will include mean, median, standard deviation, and minimum/maximum titer values at each study visit. Potential impact of anti-drug antibodies on efficacy and safety will be explored. | 1 |